CLINICAL TRIAL: NCT03162796
Title: A Phase 3, Multicenter, Randomized, Double-blind, Placebo-controlled Study Evaluating the Efficacy and Safety of Guselkumab Administered Subcutaneously in Subjects With Active Psoriatic Arthritis Including Those Previously Treated With Biologic Anti-TNF Alpha Agents
Brief Title: A Study Evaluating the Efficacy and Safety of Guselkumab Administered Subcutaneously in Participants With Active Psoriatic Arthritis Including Those Previously Treated With Biologic Anti -Tumor Necrosis Factor (TNF) Alpha Agent(s)
Acronym: Discover-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR108218; 2016-001163-37 (EudraCT Number); CNTO1959PSA3001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2017-05-19; First posted 2017-05-22 (Actual); Results first posted 2020-10-14 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-01

CONDITIONS: Arthritis, Psoriatic
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — guselkumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group 1: Guselkumab (Experimental): Participants will receive subcutaneous (SC) guselkumab 100 milligram (mg) once every 4 weeks (q4w) from Week 0 through Week 48.
  Interventions: Drug: Guselkumab
- Group 2: Guselkumab and Placebo (Experimental): Participants will receive SC guselkumab 100 mg at Weeks 0 and 4, then once every 8 weeks (q8w) (Weeks 12, 20, 28, 36, and 44) and placebo injections at other visits (Weeks 8, 16, 24, 32, 40, 48) to maintain the blind.
  Interventions: Drug: Guselkumab; Drug: Placebo
- Group 3: Placebo Followed by Guselkumab (Experimental): Participants will receive SC placebo q4w from Week 0 to Week 20, and will crossover at Week 24 to receive guselkumab 100 mg q4w from Week 24 through Week 48.
  Interventions: Drug: Guselkumab; Drug: Placebo

INTERVENTIONS:
Drug: Guselkumab — Participants will receive 100mg of guselkumab as a sterile liquid for SC injection.
  Other Names: CNTO 1959
Drug: Placebo — Participants will receive matching placebo as SC injection.
  Arms: Group 2: Guselkumab and Placebo; Group 3: Placebo Followed by Guselkumab

SUMMARY:
The primary purpose of this study is to evaluate the efficacy of guselkumab treatment in participants with active Psoriatic Arthritis (PsA) by assessing the reduction in signs and symptoms of PsA.

DETAILED DESCRIPTION:
This is a study of guselkumab in participants with active Psoriatic Arthritis (PsA) who had inadequate response to standard therapies. It will evaluate the clinical efficacy of guselkumab in the reduction of signs and symptoms and the safety profile of guselkumab in the treatment of PsA. The study will consists of 4 phases: a screening phase of up to 6 weeks, a blinded treatment phase of approximately 1 year (that is, 52 weeks), including a placebo controlled period from Week 0 to Week 24 and double-blind active treatment period from Week 24 to Week 52, and a safety follow-up phase of 8 weeks after Week 52 (Week 52 to 60) and will be 12 weeks from the last administration of study agent (at Week 48) to the final safety follow-up visit. Efficacy, safety, pharmacokinetic, immunogenicity, and biomarker evaluations will be performed in the study at defined schedule.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of Psoriatic Arthritis (PsA) for at least 6 months before the first administration of study agent and meet Classification criteria for Psoriatic Arthritis (CASPAR) at screening
* Have active PsA as defined by: at least 3 swollen joints and at least 3 tender joints at screening and at baseline; and C-reactive protein (CRP) greater than or equal to (>=) 0.3 milligram per deciLitre (mg/dL) at screening from the central laboratory
* Have at least 1 of the PsA subsets: distal interphalangeal joint involvement, polyarticular arthritis with absence of rheumatoid nodules, arthritis mutilans, asymmetric peripheral arthritis, or spondylitis with peripheral arthritis
* Have active plaque psoriasis, with at least one psoriatic plaque of >= 2 centimeter (cm) diameter or nail changes consistent with psoriasis or documented history of plaque psoriasis
* Have active PsA despite previous non-biologic disease-modifying antirheumatic drugs (DMARD), apremilast, and/or nonsteroidal anti-inflammatory drug (NSAID) therapy : Non-biologic DMARD therapy is defined as taking a non-biologic DMARD for at least 3 months or evidence of intolerance; Apremilast therapy is defined as taking apremilast at the marketed dose approved in the country where the study is being conducted for at least 4 months or evidence of intolerance; NSAID therapy is defined as taking an NSAID for at least 4 weeks or evidence of intolerance
* Participants may have been previously treated with up to 2 anti-TNF (tumor necrosis factor) alpha agents (approximately 30 percent [%] of the overall study population), and must document the reason for discontinuation

Exclusion Criteria:

* Has other inflammatory diseases that might confound the evaluations of benefit of guselkumab therapy, including but not limited to rheumatoid arthritis (RA), axial spondyloarthritis (this does not include a primary diagnosis of PsA with spondylitis), systemic lupus erythematosus, or Lyme disease
* Has ever received more than 2 anti-TNFalpha agents
* Has previously received any biologic treatment (other than anti-TNF alpha agents), including, but not limited to ustekinumab, abatacept, secukinumab, tildrakizumab, ixekizumab, brodalumab, risankizumab, or other investigative biologic treatment
* Has previously received any systemic immunosuppressants (for example, azathioprine, cyclosporine, 6 thioguanine, mercaptopurine, mycophenolate mofetil, hydroxyurea, tacrolimus) within 4 weeks of the first administration of study agent
* Has received apremilast within 4 weeks prior to the first administration of study agent
* Has previously received tofacitinib, baricitinib, filgotinib, peficitinib (ASP015K), decernotinib (VX-509), or any other Janus kinase (JAK) inhibitor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 383 (Actual)
Dates: Start 2017-08-24 (Actual); Primary Completion 2019-03-14 (Actual); Study Completion 2019-11-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (95):
- United States (9):
  - Rheumatology Associates, Birmingham, Alabama
  - Arizona Arthritis & Rheumatology Associates PC, Glendale, Arizona
  - Arizona Arthritis & Rheumatology Research, PLLC, Mesa, Arizona
  - Clinical Research Center of Connecticut, Danbury, Connecticut
  - Dawes Fretzin Clinical Research Group, LLC, Indianapolis, Indiana
  - University of Michigan, Ann Arbor, Michigan
  - Arthritis Consultants, St Louis, Missouri
  - Arthritis and Osteoporosis Associates, Freehold, New Jersey
  - Austin Regional Clinic, Austin, Texas
- Australia (6):
  - Barwon Rheumatology Services, Geelong
  - Southern Clinical Research, Hobart
  - Liverpool Hospital, Liverpool
  - Rheumatology Research Unit, Maroochydore
  - Eastern Health - Box Hill Hospital, Melbourne
  - Queen Elizabeth Hospital, Woodville South
- Canada (6):
  - Eastern Regional Health Authority, St. Clare's Mercy Hospital, St. John's, Newfoundland and Labrador
  - The Waterside Clinic, Barrie, Ontario
  - Dermatrials Research, Hamilton, Ontario
  - Skin Centre for Dermatology, Peterborough, Ontario
  - K. Papp Clinical Research, Waterloo, Ontario
  - G.R.M.O. (Groupe de recherche en maladies osseuses) Inc., Québec
- Czechia (6):
  - Revmaclinic, Brno
  - MUDr. Rosypalova, s.r.o, Ostrava
  - Revmatologicky ustav, Prague
  - Revmatologicka ambulance, Prague
  - Medical Plus S.R.O., Uherské Hradiště
  - PV-Medical S.R.O, Zlín
- Germany (5):
  - ISA GmbH, Berlin
  - Universitatsklinikum Frankfurt, Frankfurt
  - MVZ Rheuma, Hamburg
  - Rheumazentrum Ruhrgebiet, Herne
  - Krankenhaus St. Josef, Wuppertal
- Hungary (5):
  - Orszagos Reumatologia es Fizioterapias Intezet, Budapest
  - Magyar Honvedseg Egeszsegugyi Kozpont, Budapest
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - Pest Megyei Flor Ferenc Korhaz, Kistarcsa
  - Martinus Medicus Health Center, Szombathely
- Malaysia (5):
  - Hospital Selayang, Batu Caves
  - Hospital Pulau Pinang, George Town
  - Hospital Raja Permaisuri Bainun, Ipoh
  - Hospital Melaka, Malacca
  - Hospital Tuanku Jaafar, Seremban
- Poland (11):
  - Nzoz Osteo-Medic, Bialystok
  - Szpital Uniwersytecki Nr 2 w Bydgoszczy, Bydgoszcz
  - NSZOZ Unica CR, Dąbrówka
  - Centrum Kliniczno Badawcze J. Brzezicki, B. Gornikiewicz-Brzezicka Lekarze Spolka Partnerska, Elblag
  - Etyka Osrodek Badan Klinicznych, Olsztyn
  - Centrum Medyczne Hetmańska, Poznan
  - Nasz Lekarz Przychodnie Medyczne, Torun
  - Medycyna Kliniczna, Warsaw
  - Narodowy Instytut Geriatrii, Reumatologii i Rehabilitacji im. prof. dr hab. med. Eleonory Reicher, Warsaw
  - Centrum Medyczne WroMedica, Wroclaw
  - Nzoz Biogenes Sp. Z O. O., Wroclaw
- Russia (10):
  - Chelyabinsk Regional Clinical Dermatovenerological Dispensary, Chelyabinsk
  - Medical and Sanitary Unit ''Severstal'', Cherepovets
  - Krasnoyarsk State Medical University, Krasnoyarsk
  - Lipetsk Regional Dermatovenerological Dispensary, Lipetsk
  - Rostov Regional Clinical Dermatovenerological Dispensary, Rostov
  - Ryazan Regional Clinical Dermatovenerological Dispensary, Ryazan
  - Republican Clinical Hospital - G.G. Kuvatov, Ufa
  - Clinical Emergency Hospital n.a. N.V. Solovyev, Yaroslavl
  - Clinical Hospital #10, Yaroslavl
  - Research Institute of Dermatovenerology, Immunology, Yekaterinburg
- South Korea (5):
  - Seoul National University Bundang Hospital, Bundang
  - Hanyang University Hospital for rheumatic Diseases, Seoul
  - The Catholic University of Korea Seoul St. Mary's Hospital, Seoul
  - SMG - SNU Boramae Medical Center, Seoul
  - Ajou University Hospital, Suwon
- Spain (9):
  - Hosp. Univ. A Coruña, A Coruña
  - Hosp. Del Mar, Barcelona
  - Hosp. Gral. Univ. Gregorio Marañon, Madrid
  - Hosp. Univ. Ramon Y Cajal, Madrid
  - Hospital Regional Carlos Haya, Málaga
  - Hosp. Clinico Univ. de Santiago, Santiago de Compostela
  - Hosp. Infanta Luisa, Seville
  - Hosp. Unv. de Valme, Seville
  - Hosp. de Manises, Valencia
- Taiwan (8):
  - Hualien Tzu Chi Hospital, Hualien City
  - Kaohsiung Veterans General Hospital, Kaohsiung City
  - Chang Gung Memorial Hospital Kaohsiung Branch, Kaohsiung City
  - Chung Shan Medical University Hospital, Taichung
  - National Cheng Kung University Medical Center, Tainan
  - National Taiwan University Hospital, Taipei
  - Chang Kung Memorial Hospital, Taipei
  - Chang-Gung Memorial Hospital, LinKou Branch, Taoyuan District
- Ukraine (10):
  - Municipal health care institution Chernihiv Regional Hospital, Chernihiv
  - Ivano-Frankivsk National Medical University, Ivano-Frankivsk City Clinical Hospital, Ivano-Frankivsk
  - Communal Institution of Health Kharkiv City multifield hospital №18, Kharkiv
  - Municipal Institution Regional hospital-center of emergency care and disasters medicine, Kharkiv
  - Khmelnitckiy regional hospital, Khmelnytsky
  - Clinic of SI 'NSC 'The M.D.Strazhesko Institute of Cardiology' of NAMS of Ukraine', Kyiv
  - Kyiv Railway Station Clinical Hospital #2, Kyiv
  - Danylo Halytsky Lviv National Medical University, Lviv
  - Municipal Non-profit Enterprise 'Odesa Regional Clinical Hospital' Odesa Regional Council, Odesa
  - Municipal institution of Tepnopil Regional Council 'Ternopil University Hospital', Ternopil

REFERENCES:
- [Derived] Gladman DD, Eder L, Selmi C, Mease PJ, Ogdie A, Lozenski K, Adamson E, Sharaf M, Rampakakis E, Pina Vegas L, Coates LC. Influence of Biological Sex on Participant Characteristics, Guselkumab Efficacy and Radiographic Progression in Active Psoriatic Arthritis: Post Hoc Analysis of Three Randomized Trials. Rheumatol Ther. 2025 Dec 15. doi: 10.1007/s40744-025-00812-3. Online ahead of print. PMID 41396391
- [Derived] Mease P, Korotaeva T, Shesternya P, Kokhan M, Rukavitsyn A, Vasilchenkov D, Sharaf M, Lavie F, Deodhar A. Guselkumab in Biologic-Naive Patients with Active Psoriatic Arthritis in Russia: A Post Hoc Analysis of the DISCOVER-1 and -2 Randomized Clinical Trials. Rheumatol Ther. 2024 Dec;11(6):1551-1567. doi: 10.1007/s40744-024-00713-x. Epub 2024 Sep 25. PMID 39320583
- [Derived] Curtis JR, Deodhar A, Soriano ER, Rampakakis E, Shawi M, Shiff NJ, Han C, Tillett W, Gladman DD. Early Improvements with Guselkumab Associate with Sustained Control of Psoriatic Arthritis: Post hoc Analyses of Two Phase 3 Trials. Rheumatol Ther. 2024 Dec;11(6):1501-1517. doi: 10.1007/s40744-024-00702-0. Epub 2024 Sep 11. PMID 39261446
- [Derived] Baraliakos X, Gladman DD, Chakravarty SD, Gong C, Shawi M, Rampakakis E, Kishimoto M, Soriano ER, Mease PJ. BASDAI versus ASDAS in evaluating axial involvement in patients with psoriatic arthritis: a pooled analysis of two phase 3 studies. Rheumatol Adv Pract. 2024 Apr 23;8(2):rkae058. doi: 10.1093/rap/rkae058. eCollection 2024. PMID 38765190
- [Derived] Strober B, Coates LC, Lebwohl MG, Deodhar A, Leibowitz E, Rowland K, Kollmeier AP, Miller M, Wang Y, Li S, Chakravarty SD, Chan D, Shawi M, Yang YW, Thaҫi D, Rahman P. Long-Term Safety of Guselkumab in Patients with Psoriatic Disease: An Integrated Analysis of Eleven Phase II/III Clinical Studies in Psoriasis and Psoriatic Arthritis. Drug Saf. 2024 Jan;47(1):39-57. doi: 10.1007/s40264-023-01361-w. Epub 2023 Oct 31. PMID 37906417
- [Derived] Kavanaugh A, Baraliakos X, Gao S, Chen W, Sweet K, Chakravarty SD, Song Q, Shawi M, Rahman P. Genetic and Molecular Distinctions Between Axial Psoriatic Arthritis and Radiographic Axial Spondyloarthritis: Post Hoc Analyses from Four Phase 3 Clinical Trials. Adv Ther. 2023 May;40(5):2439-2456. doi: 10.1007/s12325-023-02475-4. Epub 2023 Mar 30. PMID 36995469
- [Derived] Rahman P, Boehncke WH, Mease PJ, Gottlieb AB, McInnes IB, Shawi M, Wang Y, Sheng S, Kollmeier AP, Theander E, Yu J, Leibowitz E, Marrache AM, Coates LC. Safety of Guselkumab With and Without Prior Tumor Necrosis Factor Inhibitor Treatment: Pooled Results Across 4 Studies in Patients With Psoriatic Arthritis. J Rheumatol. 2023 Jun;50(6):769-780. doi: 10.3899/jrheum.220928. Epub 2023 Jan 15. PMID 36642439
- [Derived] Orbai AM, Coates LC, Deodhar A, Helliwell PS, Ritchlin CT, Leibowitz E, Kollmeier AP, Hsia EC, Xu XL, Sheng S, Jiang Y, Liu Y, Han C. Meaningful Improvement in General Health Outcomes with Guselkumab Treatment for Psoriatic Arthritis: Patient-Reported Outcomes Measurement Information System-29 Results from a Phase 3 Study. Patient. 2022 Nov;15(6):657-668. doi: 10.1007/s40271-022-00588-6. Epub 2022 Jun 30. PMID 35768650
- [Derived] Coates LC, Ritchlin CT, Gossec L, Helliwell PS, Rahman P, Kollmeier AP, Xu XL, Shawi M, Karyekar CS, Contre C, Noel W, Sheng S, Wang Y, Xu S, Mease PJ. Guselkumab provides sustained domain-specific and comprehensive efficacy using composite indices in patients with active psoriatic arthritis. Rheumatology (Oxford). 2023 Feb 1;62(2):606-616. doi: 10.1093/rheumatology/keac375. PMID 35766811
- [Derived] Ritchlin CT, Mease PJ, Boehncke WH, Tesser J, Schiopu E, Chakravarty SD, Kollmeier AP, Xu XL, Shawi M, Jiang Y, Sheng S, Wang Y, Xu S, Merola JF, McInnes IB, Deodhar A. Sustained and improved guselkumab response in patients with active psoriatic arthritis regardless of baseline demographic and disease characteristics: pooled results through week 52 of two phase III, randomised, placebo-controlled studies. RMD Open. 2022 Mar;8(1):e002195. doi: 10.1136/rmdopen-2022-002195. PMID 35296534
- [Derived] Rahman P, Mease PJ, Helliwell PS, Deodhar A, Gossec L, Kavanaugh A, Kollmeier AP, Hsia EC, Zhou B, Lin X, Shawi M, Karyekar CS, Han C. Guselkumab demonstrated an independent treatment effect in reducing fatigue after adjustment for clinical response-results from two phase 3 clinical trials of 1120 patients with active psoriatic arthritis. Arthritis Res Ther. 2021 Jul 14;23(1):190. doi: 10.1186/s13075-021-02554-3. PMID 34261541
- [Derived] Sweet K, Song Q, Loza MJ, McInnes IB, Ma K, Leander K, Lakshminarayanan V, Franks C, Cooper P, Siebert S. Guselkumab induces robust reduction in acute phase proteins and type 17 effector cytokines in active psoriatic arthritis: results from phase 3 trials. RMD Open. 2021 May;7(2):e001679. doi: 10.1136/rmdopen-2021-001679. PMID 34011674
- [Derived] Rahman P, Ritchlin CT, Helliwell PS, Boehncke WH, Mease PJ, Gottlieb AB, Kafka S, Kollmeier AP, Hsia EC, Xu XL, Shawi M, Sheng S, Agarwal P, Zhou B, Ramachandran P, Zhuang Y, McInnes IB. Pooled Safety Results Through 1 Year of 2 Phase III Trials of Guselkumab in Patients With Psoriatic Arthritis. J Rheumatol. 2021 Dec;48(12):1815-1823. doi: 10.3899/jrheum.201532. Epub 2021 May 1. PMID 33934076
- [Derived] McGonagle D, McInnes IB, Deodhar A, Schett G, Shawi M, Kafka S, Karyekar CS, Kollmeier AP, Hsia EC, Xu XL, Sheng S, Agarwal P, Zhou B, Ritchlin CT, Rahman P, Mease PJ. Resolution of enthesitis by guselkumab and relationships to disease burden: 1-year results of two phase 3 psoriatic arthritis studies. Rheumatology (Oxford). 2021 Nov 3;60(11):5337-5350. doi: 10.1093/rheumatology/keab285. PMID 33822898
- [Derived] Deodhar A, Helliwell PS, Boehncke WH, Kollmeier AP, Hsia EC, Subramanian RA, Xu XL, Sheng S, Agarwal P, Zhou B, Zhuang Y, Ritchlin CT; DISCOVER-1 Study Group. Guselkumab in patients with active psoriatic arthritis who were biologic-naive or had previously received TNFalpha inhibitor treatment (DISCOVER-1): a double-blind, randomised, placebo-controlled phase 3 trial. Lancet. 2020 Apr 4;395(10230):1115-1125. doi: 10.1016/S0140-6736(20)30265-8. Epub 2020 Mar 13. PMID 32178765

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 383 participants were enrolled. Among them, 381 participants received at least one dose of study drug (126 in placebo group, 127 in guselkumab 100 mg q8w group and 128 in guselkumab 100 mg q4w group). One participant was randomized to guselkumab 100 mg q8w but not treated.
Pre-assignment Details: One participant was accidentally randomized before completion of screening assessments. Subsequently, this participant screen failed and was later re-screened and randomized using a new participant number.Therefore, this participant was counted twice in the number of participants enrolled, but only once in the number of participants randomized.
Groups:
- Placebo: Participants were randomized to receive placebo matched to guselkumab subcutaneous injections every 4 weeks through Week 20 in the placebo controlled period (PCP), then to receive guselkumab 100 milligrams (mg) subcutaneous injection from Week 24 every 4 weeks through Week 48 in the active treatment period.
- Guselkumab 100 mg q8w: Participants were randomized to receive guselkumab 100 mg subcutaneous injections at Weeks 0 and 4, then every 8 weeks (q8w) and placebo matched to guselkumab injections at other visits through Week 48.
- Guselkumab 100 mg q4w: Participants were randomized to receive guselkumab 100 mg subcutaneous injections every 4 weeks (q4w) through Week 48.
Period: Placebo Controlled Period: Week 0 - 24
Arm/Group | Placebo | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Started | 126 | 127 | 128
Completed | 114 | 123 | 125
Not Completed | 12 | 4 | 3
Not completed — Other | 0 | 1 | 1
Not completed — Initiated prohibited medication | 1 | 0 | 0
Not completed — Death | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 0 | 1
Not completed — Lack of Efficacy | 4 | 0 | 0
Not completed — Adverse Event | 2 | 3 | 1
Period: Active Treatment Period: Week 24 - 52
Arm/Group | Placebo | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Started | 114 | 123 | 125
Completed | 107 | 116 | 124
Not Completed | 7 | 7 | 1
Not completed — Withdrawal by Subject | 0 | 2 | 0
Not completed — Lack of Efficacy | 4 | 3 | 1
Not completed — Adverse Event | 3 | 2 | 0
Period: Safety Follow-up: Week 52 - 60
Arm/Group | Placebo | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Started | 107 | 116 | 124
Completed | 106 | 114 | 123
Not Completed | 1 | 2 | 1
Not completed — Withdrawal by Subject | 1 | 2 | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) 1 included all participants who received at least 1 dose (complete/partial) of study agent according to randomized treatment group regardless of treatment actually received.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w | Total
Number analyzed (Participants) | 126 | 127 | 128 | 381
Age, Continuous [Mean (Standard Deviation); unit: years] | 49 (11.1) | 48.9 (11.52) | 47.4 (11.59) | 48.4 (11.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 59 | 62 | 186
  Male | 61 | 68 | 66 | 195
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 0 | 4
  Not Hispanic or Latino | 122 | 124 | 128 | 374
  Unknown or Not Reported | 2 | 1 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 12 | 10 | 7 | 29
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Black or African American | 0 | 0 | 0 | 0
  White | 112 | 116 | 121 | 349
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 0 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  AUSTRALIA | 5 | 8 | 4 | 17
  CANADA | 8 | 3 | 4 | 15
  CZECH REPUBLIC | 5 | 4 | 3 | 12
  GERMANY | 3 | 10 | 10 | 23
  HUNGARY | 3 | 4 | 9 | 16
  MALAYSIA | 5 | 1 | 2 | 8
  POLAND | 37 | 36 | 34 | 107
  RUSSIAN FEDERATION | 22 | 19 | 23 | 64
  SOUTH KOREA | 3 | 1 | 0 | 4
  SPAIN | 5 | 6 | 1 | 12
  TAIWAN | 4 | 7 | 5 | 16
  UKRAINE | 19 | 22 | 29 | 70
  UNITED STATES | 7 | 6 | 4 | 17

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved an American College of Rheumatology (ACR) 20 Response at Week 24
Description: ACR 20 response: >=20% improvement from baseline in both swollen joint count (66 joints) and tender joint count (68 joints), and >=20% improvement from baseline in 3 of 5 assessments: patient's assessment of pain using visual analog scale (VAS; 0-100 mm, 0=no pain and 100=worst possible pain), patient's global assessment of disease activity (arthritis, VAS; 0-100 mm, 0=excellent and 100= poor), physician's global assessment of disease activity (VAS; 0-100 mm, 0=no arthritis activity and 100=extremely active arthritis), patient's assessment of physical function measured by Disability Index of Health Assessment Questionnaire (HAQ-DI; 20-question instrument assessing 8 functional areas; range: 0-3, 0= no difficulty, 3= inability to perform task in that area), and CRP. Treatment Failure (TF) criteria- discontinued study drug, initiated/increased dose of non-biologic disease-modifying antirheumatic drugs (DMARDs) or oral corticosteroids, initiated prohibited psoriatic arthritis treatment.
Time Frame: Week 24
Population: Analysis population is full analysis set 1 (FAS1). Participants who achieved ACR 20 response at Week 24 and did not meet any TF criteria before Week 24 were considered as responders. Participants who met 1 or more TF criteria or with missing data were considered as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 126 | 127 | 128
percentage of participants | 22.2 | 52.0 | 59.4
Statistical Analysis 1: Comparison: Placebo vs Guselkumab 100 mg q8w; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Difference in percentage = 29.8, 95% CI 2-sided [18.6 to 41.1]
Statistical Analysis 2: Comparison: Placebo vs Guselkumab 100 mg q4w; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Difference in percentage = 37.1, 95% CI 2-sided [26.1 to 48.2]

2. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire-Disability Index (HAQ-DI) Score at Week 24
Description: HAQ-DI score assess functional status of participant. It is 20 question instrument that assess degree of difficulty a person has in accomplishing tasks in 8 functional areas (dressing, arising, eating, walking, hygiene, reaching, gripping, and activities of daily living). Responses in each functional area were scored from 0=indicating no difficulty, to 3=indicating inability to perform a task in that area. Total HAQ score is average of the computed categories scores ranging from 0-3 where 0=least difficulty and 3=extreme difficulty. Lower scores are indicative of better functioning. Negative change from baseline indicates improvement of physical function.
Time Frame: Baseline and Week 24
Population: Analysis population is FAS1. Data after meeting one or more TF criteria were imputed as no change from baseline. Missing data were assumed to be missing at random (MAR) and imputed using multiple imputation (MI).
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 126 | 127 | 128
units on a scale | -0.0743 [-0.1605 to 0.0119] | -0.3225 [-0.4082 to -0.2369] | -0.3968 [-0.4825 to -0.3112]
Statistical Analysis 1: Comparison: Placebo vs Guselkumab 100 mg q8w; Test type: Superiority; p < 0.001, ANCOVA; Least Square (LS) Mean Difference = -0.2483, 95% CI 2-sided [-0.3640 to -0.1325]
Statistical Analysis 2: Comparison: Placebo vs Guselkumab 100 mg q4w; Test type: Superiority; p < 0.001, ANCOVA; LS Mean difference = -0.3226, 95% CI 2-sided [-0.4385 to -0.2066]

3. Secondary Outcome: Percentage of Participants Who Achieved an American College of Rheumatology (ACR) 50 Response at Week 24
Description: ACR 50 response was defined as greater than or equal to (>=)50 percent (%) improvement from baseline in both swollen joint count (66 joints) and tender joint count (68 joints), and >=50% improvement from baseline in 3 of 5 assessments: patient's assessment of pain using visual analog scale (VAS; 0-100 mm, 0=no pain and 100=worst possible pain), patient's global assessment of disease activity (arthritis, VAS; 0-100 mm, 0=excellent and 100= poor), physician's global assessment of disease activity (VAS; 0-100 mm, 0=no arthritis activity and 100=extremely active arthritis), patient's assessment of physical function measured by Disability Index of the Health Assessment Questionnaire (HAQ-DI; a 20-question instrument assessing 8 functional areas; range: 0-3, 0=no difficulty, 3=inability to perform a task in that area), and C-Reactive Protein (CRP).
Time Frame: Week 24
Population: Analysis population is FAS1. Participants who achieved ACR 50 response at Week 24 and did not meet any TF criteria before Week 24 were considered as responders. Participants who met 1 or more TF criteria or with missing data were considered as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 126 | 127 | 128
percentage of participants | 8.7 | 29.9 | 35.9
Statistical Analysis 1: Comparison: Placebo vs Guselkumab 100 mg q8w; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — Nominal; Difference in percentage = 21.4, 95% CI 2-sided [12.1 to 30.7]
Statistical Analysis 2: Comparison: Placebo vs Guselkumab 100 mg q4w; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — Nominal; Difference in percentage = 27.2, 95% CI 2-sided [17.6 to 36.8]

4. Secondary Outcome: Percentage of Participants With Psoriasis Response of IGA (Score: 0[Cleared] or 1[Minimal] and >=2 Grade Reduction From Baseline) at Week 24 Among Participants With >=3% Body Surface Area (BSA) Psoriatic Involvement and IGA Score of >=2 (Mild) at Baseline
Description: A psoriasis Investigator's Global Assessment (IGA) response was defined as an IGA score of 0 (cleared) or 1 (minimal) and >=2 grade reduction from baseline in the IGA psoriasis score. The IGA documents the investigator's assessment of the patient's psoriasis and lesions are graded for induration, erythema and scaling, each using a 5 point scale: 0 (no evidence), 1 (minimal), 2 (mild), 3 (moderate), and 4 (severe). The IGA score of psoriasis was based upon the average of induration, erythema and scaling scores. The participant's psoriasis was assessed as cleared (0), minimal (1), mild (2), moderate (3), or severe (4).
Time Frame: Week 24
Population: FAS1 among the participants with >=3% BSA psoriatic involvement and an IGA score of >=2 (mild) at baseline. Participants who achieved psoriasis IGA response at Week 24 and did not meet any TF criteria before Week 24 were considered as responders. Participants who met 1 or more TF criteria or with missing data were considered as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 78 | 82 | 89
percentage of participants | 15.4 | 57.3 | 75.3
Statistical Analysis 1: Comparison: Placebo vs Guselkumab 100 mg q8w; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Difference in percentage = 42.0, 95% CI 2-sided [28.9 to 55.1]
Statistical Analysis 2: Comparison: Placebo vs Guselkumab 100 mg q4w; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Difference in percentage = 60.0, 95% CI 2-sided [48.3 to 71.8]

5. Secondary Outcome: Percentage of Participants Who Achieved an American College of Rheumatology (ACR) 20 Response at Week 16
Description: ACR 20 response: >=20% improvement from baseline in both swollen joint count (66 joints) and tender joint count (68 joints), and >=20% improvement from baseline in 3 of 5 assessments: patient's assessment of pain using visual analog scale (VAS; 0-100 mm, 0=no pain and 100=worst possible pain), patient's global assessment of disease activity (arthritis, VAS; 0-100 mm, 0=excellent and 100= poor), physician's global assessment of disease activity (VAS; 0-100 mm, 0=no arthritis activity and 100=extremely active arthritis), patient's assessment of physical function measured by Disability Index of Health Assessment Questionnaire (HAQ-DI; 20-question instrument assessing 8 functional areas; range: 0-3, 0=indicating no difficulty, 3=indicating inability to perform task in that area), and C-reactive protein (CRP).
Time Frame: Week 16
Population: Analysis population is FAS1. Participants who achieved ACR 20 response at Week 16 and did not meet any TF criteria before Week 16 were considered as responders. Participants who met 1 or more TF criteria or with missing data were considered as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 126 | 127 | 128
percentage of participants | 25.4 | 52.0 | 60.2
Statistical Analysis 1: Comparison: Placebo vs Guselkumab 100 mg q8w; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — Nominal; Difference in percentage = 26.7, 95% CI 2-sided [15.3 to 38.1]
Statistical Analysis 2: Comparison: Placebo vs Guselkumab 100 mg q4w; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — Nominal; Difference in percentage = 34.8, 95% CI 2-sided [23.5 to 46.0]

6. Secondary Outcome: Change From Baseline in Disease Activity Score (DAS28) (C-reactive Protein [CRP]) Score at Week 24
Description: The Disease Activity Index Score (DAS28) based on C-Reactive Protein (CRP) is an index combining tender joints (28 joints), swollen joints (28 joints), CRP and patient's global assessment of disease activity. The set of 28 joint count is based on evaluation of the shoulder, elbow, wrist, metacarpophalangeal (MCP) MCP1 to MCP5, proximal interphalangeal (PIP) PIP1 to PIP5 joints of both the upper right extremity and the upper left extremity as well as the knee joints of lower right and lower left extremities. The values are 0=best to 10=worst. Negative changes from baseline indicate improvement of arthritis.
Time Frame: Baseline and Week 24
Population: Analysis population is FAS1. Data after meeting one or more TF criteria were imputed as no change from baseline. Missing data were assumed to be MAR and imputed using MI.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 126 | 127 | 128
units on a scale | -0.70 [-0.89 to -0.51] | -1.43 [-1.61 to -1.24] | -1.61 [-1.80 to -1.42]
Statistical Analysis 1: Comparison: Placebo vs Guselkumab 100 mg q8w; Test type: Superiority; p < 0.001, ANCOVA — Nominal; LS Mean difference = -0.73, 95% CI [-0.98 to -0.48]
Statistical Analysis 2: Comparison: Placebo vs Guselkumab 100 mg q4w; Test type: Superiority; p < 0.001, ANCOVA — Nominal; LS Mean difference = -0.91, 95% CI [-1.16 to -0.66]

7. Secondary Outcome: Percentage of Participants Who Achieve an American College of Rheumatology (ACR) 70 Response at Week 24
Description: ACR 70 response was defined as >= 70% improvement from baseline in both swollen joint count (66 joints) and tender joint count (68 joints), and >=70% improvement from baseline in 3 of 5 assessments: patient's assessment of pain using visual analog scale (VAS; 0-100 mm, 0=no pain and 100=worst possible pain), patient's global assessment of disease activity (arthritis, VAS; 0-100 mm, 0=excellent and 100= poor), physician's global assessment of disease activity (VAS; 0-100 mm, 0=no arthritis activity and 100=extremely active arthritis), patient's assessment of physical function measured by Disability Index of the Health Assessment Questionnaire (HAQ-DI; a 20-question instrument assessing 8 functional areas; range: 0-3, 0=no difficulty, 3=inability to perform a task in that area), and CRP.
Time Frame: Week 24
Population: Analysis population is FAS1. Participants who achieved ACR 70 response at Week 24 and did not meet any TF criteria before Week 24 were considered as responders. Participants who met 1 or more TF criteria or with missing data were considered as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 126 | 127 | 128
percentage of participants | 5.6 | 11.8 | 20.3
Statistical Analysis 1: Comparison: Placebo vs Guselkumab 100 mg q8w; Test type: Superiority; p = 0.069, Cochran-Mantel-Haenszel; Difference in percentage = 6.4, 95% CI 2-sided [-0.3 to 13.1]
Statistical Analysis 2: Comparison: Placebo vs Guselkumab 100 mg q4w; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Difference in percentage = 14.8, 95% CI 2-sided [6.9 to 22.7]

8. Secondary Outcome: Percentage of Participants Who Achieved an American College of Rheumatology (ACR) 50 Response at Week 16
Description: ACR 50 response was defined as >=50% improvement from baseline in both swollen joint count (66 joints) and tender joint count (68 joints), and >=50% improvement from baseline in 3 of 5 assessments: patient's assessment of pain using visual analog scale (VAS; 0-100 mm, 0=no pain and 100=worst possible pain), patient's global assessment of disease activity (arthritis, VAS; 0-100 mm, 0=excellent and 100= poor), physician's global assessment of disease activity (VAS; 0-100 mm, 0=no arthritis activity and 100=extremely active arthritis), patient's assessment of physical function measured by Disability Index of the Health Assessment Questionnaire (HAQ-DI; a 20-question instrument assessing 8 functional areas; range: 0-3, 0=no difficulty, 3=inability to perform a task in that area), and CRP.
Time Frame: Week 16
Population: Analysis population is FAS1. Participants who achieved ACR 50 response at Week 16 and did not meet any TF criteria before Week 16 were considered as responders. Participants who met 1 or more TF criteria or with missing data were considered as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 126 | 127 | 128
percentage of participants | 12.7 | 22.8 | 26.6
Statistical Analysis 1: Comparison: Placebo vs Guselkumab 100 mg q8w; Test type: Superiority; p = 0.036, Cochran-Mantel-Haenszel — Nominal; Difference in percentage = 10.2, 95% CI 2-sided [1.0 to 19.3]
Statistical Analysis 2: Comparison: Placebo vs Guselkumab 100 mg q4w; Test type: Superiority; p = 0.006, Cochran-Mantel-Haenszel — Nominal; Difference in percentage = 13.9, 95% CI 2-sided [4.4 to 23.4]

9. Secondary Outcome: Change From Baseline in 36-Item Short Form Health Survey (SF-36) Physical Component Summary (PCS) Score at Week 24
Description: SF-36 is a multi-domain instrument with 36 items to evaluate the health status and quality of life. It included 8 subscales (physical functioning, physical role functioning, bodily pain, general health perception, vitality, social functioning, emotional role functioning, and mental health), which yielded a Physical Component Summary (PCS) with score range 0-100 (higher score-better quality of life) and a Mental Component Summary (MCS) with score range 0-100 (higher score-better quality of life) in addition to subscale scores. The PCS scores are normalized to a mean of 50 and standard deviations of 10, based upon general US population norms. A positive change indicates improvement while a negative change indicates worsening of health status and quality of life.
Time Frame: Baseline and Week 24
Population: as for outcome 6
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 126 | 127 | 128
units on a scale | 1.96 [0.69 to 3.24] | 6.10 [4.83 to 7.37] | 6.87 [5.60 to 8.14]
Statistical Analysis 1: Comparison: Placebo vs Guselkumab 100 mg q8w; Test type: Superiority; p < 0.001, ANCOVA; LS Mean difference = 4.14, 95% CI 2-sided [2.42 to 5.85]
Statistical Analysis 2: Comparison: Placebo vs Guselkumab 100 mg q4w; Test type: Superiority; p < 0.001, ANCOVA; LS Mean difference = 4.91, 95% CI [3.19 to 6.63]

10. Secondary Outcome: Percentage of Participants With Resolution of Enthesitis at Week 24 Among the Participants With Enthesitis at Baseline
Description: Enthesitis was assessed using the Leeds Enthesitis Index (LEI), a tool developed to assess enthesitis in participants with PsA and evaluates the presence (score of 1) or absence (score of 0) of pain by applying local pressure to the following entheses: left and right lateral epicondyle humerus, left and right medial femoral condyle, and left and right achilles tendon insertion. The enthesitis index score is a total score of the 6 evaluated sites from 0 (0 sites with tenderness) to 6 (worst possible score; 6 sites with tenderness). A LEI score of 0 at a post baseline visit indicates resolution of enthesitis when baseline LEI greater than (>) 0.
Time Frame: Week 24
Population: Analysis population is FAS1 among the participants with enthesitis (LEI) at baseline. Participants who achieved resolution of enthesitis at Week 24 and did not meet any TF criteria before Week 24 were considered as responders. Participants who met 1 or more TF criteria or with missing data were considered as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 77 | 72 | 73
percentage of participants | 27.3 | 40.3 | 47.9
Statistical Analysis 1: Comparison: Placebo vs Guselkumab 100 mg q8w; Test type: Superiority; p = 0.094, Cochran-Mantel-Haenszel — Nominal; Difference in percentage = 13.0, 95% CI 2-sided [-1.6 to 27.5]
Statistical Analysis 2: Comparison: Placebo vs Guselkumab 100 mg q4w; Test type: Superiority; p = 0.013, Cochran-Mantel-Haenszel — Nominal; Difference in percentage = 19.8, 95% CI 2-sided [4.9 to 34.6]

11. Secondary Outcome: Change From Baseline in Enthesitis Score (Based on LEI) at Week 24 Among the Participants With Enthesitis at Baseline
Description: Enthesitis was assessed using the LEI, a tool developed to assess enthesitis in participants with PsA and evaluates the presence (score of 1) or absence (score of 0) of pain by applying local pressure to the following entheses: left and right lateral epicondyle humerus, left and right medial femoral condyle, and left and right achilles tendon insertion. The enthesitis index score is a total score of the 6 evaluated sites from 0 (0 sites with tenderness) to 6 (worst possible score; 6 sites with tenderness). Negative changes from baseline indicates improvement of enthesitis.
Time Frame: Baseline and Week 24
Population: Analysis population is FAS1 among the participants with enthesitis (LEI) at baseline. Data after meeting one or more TF criteria were imputed as no change from baseline. Missing data were assumed to be MAR and imputed using MI.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 77 | 72 | 73
units on a scale | -1.01 [-1.37 to -0.66] | -1.35 [-1.72 to -0.98] | -1.75 [-2.13 to -1.38]
Statistical Analysis 1: Comparison: Placebo vs Guselkumab 100 mg q8w; Test type: Superiority; p = 0.185, ANCOVA — Nominal; LS Mean difference = -0.33, 95% CI 2-sided [-0.83 to 0.16]
Statistical Analysis 2: Comparison: Placebo vs Guselkumab 100 mg q4w; Test type: Superiority; p = 0.004, ANCOVA — Nominal; LS Mean difference = -0.74, 95% CI 2-sided [-1.24 to -0.24]

12. Secondary Outcome: Change From Baseline in 36-Item Short Form Health Survey (SF-36) Mental Component Summary (MCS) Score at Week 24
Description: SF-36 is a multi-domain instrument with 36 items to evaluate the health status and quality of life. It included 8 subscales (physical functioning, physical role functioning, bodily pain, general health perception, vitality, social functioning, emotional role functioning, and mental health), which yielded a Physical Component Summary (PCS) with score range 0-100 (higher score-better quality of life) and a Mental Component Summary (MCS) with score range 0-100 (higher score-better quality of life) in addition to subscale scores. The MCS scores are normalized to a mean of 50 and standard deviations of 10, based upon general US population norms. A positive change indicates improvement while a negative change indicates worsening of health status and quality of life.
Time Frame: Baseline and Week 24
Population: as for outcome 6
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 126 | 127 | 128
units on a scale | 2.37 [0.93 to 3.81] | 3.20 [1.78 to 4.63] | 3.60 [2.17 to 5.02]
Statistical Analysis 1: Comparison: Placebo vs Guselkumab 100 mg q8w; Test type: Superiority; p = 0.398, ANCOVA — Nominal; LS Mean difference = 0.83, 95% CI 2-sided [-1.10 to 2.77]
Statistical Analysis 2: Comparison: Placebo vs Guselkumab 100 mg q4w; Test type: Superiority; p = 0.214, ANCOVA — Nominal; LS Mean difference = 1.23, 95% CI 2-sided [-0.71 to 3.16]

13. Secondary Outcome: Percentage of Participants With Resolution of Dactylitis at Week 24 Among the Participants With Dactylitis at Baseline
Description: The presence and severity of dactylitis was assessed in both hands and feet using a scoring system from 0 to 3 (0-no dactylitis, 1-mild dactylitis, 2-moderate dactylitis, and 3-severe dactylitis) for each digit. The results were summed to produce a final score ranging from 0 to 60. Higher score indicates more severe dactylitis. Resolution of dactylitis was defined as a dactylitis score of 0 with the baseline dactylitis score >0.
Time Frame: Week 24
Population: Analysis population is FAS1 among the participants with dactylitis at baseline. Participants who achieved resolution of dactylitis at Week 24 and did not meet any TF criteria before Week 24 were considered as responders. Participants who met 1 or more TF criteria or with missing data were considered as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 55 | 49 | 38
percentage of participants | 49.1 | 65.3 | 63.2
Statistical Analysis 1: Comparison: Placebo vs Guselkumab 100 mg q8w; Test type: Superiority; p = 0.088, Cochran-Mantel-Haenszel — Nominal; Difference in percentage = 16.6, 95% CI 2-sided [-1.5 to 34.8]
Statistical Analysis 2: Comparison: Placebo vs Guselkumab 100 mg q4w; Test type: Superiority; p = 0.212, Cochran-Mantel-Haenszel — Nominal; Difference in percentage = 13.4, 95% CI 2-sided [-6.9 to 33.7]

14. Secondary Outcome: Change From Baseline in Dactylitis Scores at Week 24 Among the Participants With Dactylitis at Baseline
Description: The presence and severity of dactylitis was assessed in both hands and feet using a scoring system from 0 to 3 (0-no dactylitis, 1-mild dactylitis, 2-moderate dactylitis, and 3-severe dactylitis) for each digit. The results were summed to produce a final score ranging from 0 to 60. A higher score indicates more severe dactylitis. Negative change from baseline indicates improvement in dactylitis.
Time Frame: Baseline and Week 24
Population: Analysis population is FAS1 among the participants with dactylitis at baseline. Data after meeting one or more TF criteria were imputed as no change from baseline. Missing data were assumed to be MAR and imputed using MI.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 55 | 49 | 38
units on a scale | -4.30 [-5.96 to -2.63] | -6.11 [-7.81 to -4.41] | -5.82 [-7.82 to -3.83]
Statistical Analysis 1: Comparison: Placebo vs Guselkumab 100 mg q8w; Test type: Superiority; p = 0.121, ANCOVA — Nominal; LS Mean difference = -1.82, 95% CI 2-sided [-4.12 to 0.49]
Statistical Analysis 2: Comparison: Placebo vs Guselkumab 100 mg q4w; Test type: Superiority; p = 0.225, ANCOVA — Nominal; LS Mean difference = -1.53, 95% CI 2-sided [-4.00 to 0.95]

15. Secondary Outcome: Percentage of Participants Who Achieved ACR 20 Response by Visit Over Time Through Week 24
Description: ACR 20 response was defined as >=20% improvement from baseline in both swollen joint count (66 joints) and tender joint count (68 joints), and >=20% improvement from baseline in 3 of the 5 assessments: patient's assessment of pain using VAS (0-100 mm, 0=no pain and 100=worst possible pain), patient's global assessment of disease activity (arthritis, VAS; 0-100 mm, 0=excellent and 100= poor), physician's global assessment of disease activity (VAS; 0-100 mm, 0=no arthritis activity and 100=extremely active arthritis), patient's assessment of physical function measured by HAQ-DI (defined as a 20-question instrument assessing 8 functional areas; range: 0-3, 0=indicating no difficulty, 3=indicating inability to perform a task in that area), and CRP.
Time Frame: Weeks 4, 8, 12, 16, 20 and 24
Population: Analysis population is FAS1. Participants who achieved ACR 20 response at a specific time point and did not meet any treatment failure (TF) criteria before, were considered as responders at that time point. Participants who met 1 or more TF criteria before or with missing data at that time point were considered as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 126 | 127 | 128
percentage of participants
  Week 4 | 7.9 | 15.7 | 20.3
  Week 8 | 18.3 | 36.2 | 39.1
  Week 12 | 27.0 | 43.3 | 53.1
  Week 16 | 25.4 | 52.0 | 60.2
  Week 20 | 30.2 | 51.2 | 62.5
  Week 24 | 22.2 | 52.0 | 59.4

16. Secondary Outcome: Percentage of Participants Who Achieved ACR 50 Response by Visit Over Time Through Week 24
Description: ACR 50 response was defined as >=50% improvement from baseline in both swollen joint count (66 joints) and tender joint count (68 joints), and >=50% improvement from baseline in 3 of the 5 assessments: patient's assessment of pain using VAS (0-100 mm, 0=no pain and 100=worst possible pain), patient's global assessment of disease activity (arthritis, VAS; 0-100 mm, 0=excellent and 100= poor), physician's global assessment of disease activity (VAS; 0-100 mm, 0=no arthritis activity and 100=extremely active arthritis), patient's assessment of physical function measured by HAQ-DI (defined as a 20-question instrument assessing 8 functional areas; range: 0-3, 0=indicating no difficulty, 3=indicating inability to perform a task in that area), and CRP.
Time Frame: Weeks 4, 8, 12, 16, 20 and 24
Population: Analysis population is FAS1. Participants who achieved ACR 50 response at a specific time point and did not meet any treatment failure (TF) criteria before, were considered as responders at that time point. Participants who met 1 or more TF criteria before or with missing data at that time point were considered as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 126 | 127 | 128
percentage of participants
  Week 4 | 2.4 | 1.6 | 3.1
  Week 8 | 7.9 | 7.9 | 10.9
  Week 12 | 10.3 | 20.5 | 24.2
  Week 16 | 12.7 | 22.8 | 26.6
  Week 20 | 13.5 | 29.1 | 37.5
  Week 24 | 8.7 | 29.9 | 35.9

17. Secondary Outcome: Percentage of Participants Who Achieved ACR 70 Response by Visit Over Time Through Week 24
Description: ACR 70 response was defined as >=70% improvement from baseline in both swollen joint count (66 joints) and tender joint count (68 joints), and >=70% improvement from baseline in 3 of the 5 assessments: patient's assessment of pain using VAS (0-100 millimeters [mm], 0=no pain and 100=worst possible pain), patient's global assessment of disease activity (arthritis, VAS; 0-100 mm, 0=excellent and 100= poor), physician's global assessment of disease activity (VAS; 0-100 mm, 0=no arthritis activity and 100=extremely active arthritis), patient's assessment of physical function measured by HAQ-DI (defined as a 20-question instrument assessing 8 functional areas; range: 0-3, 0=indicating no difficulty, 3=indicating inability to perform a task in that area), and CRP.
Time Frame: Weeks 4, 8, 12, 16, 20 and 24
Population: Analysis population is FAS1. Participants who achieved ACR 70 response at a specific time point and did not meet any TF criteria before, were considered as responders at that time point. Participants who met 1 or more TF criteria before or with missing data at that time point were considered as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 126 | 127 | 128
percentage of participants
  Week 4 | 0 | 0.8 | 0
  Week 8 | 1.6 | 3.1 | 2.3
  Week 12 | 4.8 | 7.1 | 6.3
  Week 16 | 5.6 | 7.9 | 7.8
  Week 20 | 7.1 | 11.8 | 17.2
  Week 24 | 5.6 | 11.8 | 20.3

18. Secondary Outcome: ACR Components- Swollen Joint Count and Tender Joint Count Through Week 24
Description: ACR components including swollen joint count (66 joints) and tender joint count (68 joints) were measured.
Time Frame: Weeks 4, 8, 12, 16, 20 and 24
Population: Analysis population is FAS1. Here, n (number analyzed) signifies the number of participants analyzed at specified timepoints.
Measure: Mean (Standard Deviation); unit: joints
Arm/Group | Placebo | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 126 | 127 | 128
joints
  Week 4: Swollen Joint Count: number analyzed (Participants) | 124 | 124 | 128
  Week 4: Swollen Joint Count | 8.0 (7.71) | 7.7 (7.89) | 5.7 (4.89)
  Week 8: Swollen Joint Count: number analyzed (Participants) | 122 | 125 | 128
  Week 8: Swollen Joint Count | 6.6 (5.83) | 6.2 (9.36) | 4.4 (5.22)
  Week 12: Swollen Joint Count: number analyzed (Participants) | 123 | 126 | 127
  Week 12: Swollen Joint Count | 6.1 (6.41) | 4.5 (6.63) | 3.5 (5.60)
  Week 16: Swollen Joint Count: number analyzed (Participants) | 122 | 123 | 127
  Week 16: Swollen Joint Count | 5.9 (6.09) | 3.8 (5.15) | 2.7 (4.25)
  Week 20: Swollen Joint Count: number analyzed (Participants) | 118 | 122 | 126
  Week 20: Swollen Joint Count | 5.2 (5.72) | 4.0 (6.28) | 2.7 (4.87)
  Week 24: Swollen Joint Count: number analyzed (Participants) | 118 | 123 | 127
  Week 24: Swollen Joint Count | 4.9 (6.14) | 3.8 (6.53) | 2.8 (5.27)
  Week 4: Tender Joint Count: number analyzed (Participants) | 124 | 124 | 128
  Week 4: Tender Joint Count | 17.0 (13.81) | 16.3 (14.11) | 14.4 (11.85)
  Week 8: Tender Joint Count: number analyzed (Participants) | 122 | 125 | 128
  Week 8: Tender Joint Count | 15.8 (13.68) | 13.5 (13.86) | 12.2 (11.53)
  Week 12: Tender Joint Count: number analyzed (Participants) | 123 | 126 | 127
  Week 12: Tender Joint Count | 15.1 (14.21) | 11.5 (13.16) | 9.7 (11.14)
  Week 16: Tender Joint Count: number analyzed (Participants) | 122 | 123 | 127
  Week 16: Tender Joint Count | 15.5 (13.61) | 10.3 (12.06) | 9.0 (10.29)
  Week 20: Tender Joint Count: number analyzed (Participants) | 118 | 122 | 126
  Week 20: Tender Joint Count | 13.4 (13.02) | 9.9 (12.53) | 7.9 (9.54)
  Week 24: Tender Joint Count: number analyzed (Participants) | 118 | 123 | 127
  Week 24: Tender Joint Count | 13.2 (12.09) | 9.9 (12.82) | 8.4 (10.47)

19. Secondary Outcome: ACR Components- Patient's Assessment of Pain, Patient's Global Assessment of Disease Activity, Physician's Global Assessment of Disease Activity Through Week 24
Description: ACR components included patient's assessment of pain using visual analog scale (VAS; 0-100 mm, 0=no pain and 100=worst possible pain), patient's global assessment (PtGA) of disease activity (arthritis, VAS; 0-100 mm, 0=excellent and 100= poor), physician's global assessment (PGA) of disease activity (VAS; 0-100 mm, 0=no arthritis activity and 100=extremely active arthritis).
Time Frame: Weeks 4, 8, 12, 16, 20 and 24
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Placebo | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 126 | 127 | 128
millimeters
  Week 4: Patient's Assessment of Pain: number analyzed (Participants) | 124 | 123 | 128
  Week 4: Patient's Assessment of Pain | 5.74 (2.296) | 5.49 (2.159) | 5.18 (2.224)
  Week 8: Patient's Assessment of Pain: number analyzed (Participants) | 123 | 126 | 128
  Week 8: Patient's Assessment of Pain | 5.06 (2.257) | 4.90 (2.310) | 4.54 (2.397)
  Week 12: Patient's Assessment of Pain: number analyzed (Participants) | 123 | 126 | 127
  Week 12: Patient's Assessment of Pain | 4.96 (2.355) | 4.35 (2.503) | 4.09 (2.346)
  Week 16: Patient's Assessment of Pain: number analyzed (Participants) | 122 | 124 | 127
  Week 16: Patient's Assessment of Pain | 5.01 (2.417) | 4.25 (2.471) | 3.85 (2.462)
  Week 20: Patient's Assessment of Pain: number analyzed (Participants) | 118 | 124 | 126
  Week 20: Patient's Assessment of Pain | 4.98 (2.497) | 4.00 (2.481) | 3.51 (2.409)
  Week 24: Patient's Assessment of Pain: number analyzed (Participants) | 118 | 123 | 127
  Week 24: Patient's Assessment of Pain | 5.09 (2.379) | 3.82 (2.470) | 3.52 (2.502)
  Week 4: PtGA of Disease Activity: number analyzed (Participants) | 124 | 123 | 128
  Week 4: PtGA of Disease Activity | 5.86 (2.281) | 5.80 (2.181) | 5.36 (2.200)
  Week 8: PtGA of Disease Activity: number analyzed (Participants) | 123 | 126 | 128
  Week 8: PtGA of Disease Activity | 5.26 (2.271) | 4.99 (2.381) | 4.82 (2.384)
  Week 12: PtGA of Disease Activity: number analyzed (Participants) | 123 | 126 | 127
  Week 12: PtGA of Disease Activity | 5.13 (2.398) | 4.46 (2.459) | 4.18 (2.441)
  Week 16: PtGA of Disease Activity: number analyzed (Participants) | 122 | 124 | 127
  Week 16: PtGA of Disease Activity | 5.12 (2.379) | 4.59 (2.541) | 3.96 (2.458)
  Week 20: PtGA of Disease Activity: number analyzed (Participants) | 118 | 124 | 126
  Week 20: PtGA of Disease Activity | 5.08 (2.596) | 4.21 (2.604) | 3.57 (2.443)
  Week 24: PtGA of Disease Activity: number analyzed (Participants) | 118 | 123 | 127
  Week 24: PtGA of Disease Activity | 5.19 (2.419) | 4.03 (2.603) | 3.48 (2.412)
  Week 4: PGA of Disease Activity: number analyzed (Participants) | 122 | 123 | 126
  Week 4: PGA of Disease Activity | 5.53 (1.986) | 4.94 (1.977) | 4.72 (1.955)
  Week 8: PGA of Disease Activity: number analyzed (Participants) | 122 | 125 | 128
  Week 8: PGA of Disease Activity | 4.79 (2.197) | 3.88 (2.299) | 3.63 (2.035)
  Week 12: PGA of Disease Activity: number analyzed (Participants) | 122 | 125 | 127
  Week 12: PGA of Disease Activity | 4.31 (2.196) | 3.47 (1.992) | 3.08 (2.031)
  Week 16: PGA of Disease Activity: number analyzed (Participants) | 120 | 123 | 124
  Week 16: PGA of Disease Activity | 4.31 (2.296) | 3.39 (2.260) | 2.73 (2.022)
  Week 20: PGA of Disease Activity: number analyzed (Participants) | 117 | 121 | 125
  Week 20: PGA of Disease Activity | 3.96 (2.367) | 2.90 (2.132) | 2.44 (1.780)
  Week 24: PGA of Disease Activity: number analyzed (Participants) | 117 | 122 | 127
  Week 24: PGA of Disease Activity | 4.07 (2.361) | 2.81 (2.169) | 2.34 (1.889)

20. Secondary Outcome: ACR Component- C-reactive Protein (CRP) Through Week 24
Description: ACR component including CRP was measured.
Time Frame: Weeks 4, 8, 12, 16, 20 and 24
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: milligrams per deciliter (mg/dL)
Arm/Group | Placebo | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 126 | 127 | 128
milligrams per deciliter (mg/dL)
  Week 4: number analyzed (Participants) | 124 | 123 | 128
  Week 4 | 1.220 (1.5753) | 1.159 (1.7641) | 0.785 (1.1917)
  Week 8: number analyzed (Participants) | 120 | 124 | 127
  Week 8 | 1.184 (1.8722) | 1.059 (1.4736) | 0.720 (1.2637)
  Week 12: number analyzed (Participants) | 122 | 123 | 127
  Week 12 | 1.138 (1.5889) | 0.936 (1.3470) | 0.629 (0.7882)
  Week 16: number analyzed (Participants) | 120 | 123 | 124
  Week 16 | 1.143 (1.6005) | 0.996 (1.5296) | 0.592 (0.7861)
  Week 20: number analyzed (Participants) | 119 | 124 | 126
  Week 20 | 1.105 (1.6401) | 0.941 (1.5067) | 0.592 (0.8831)
  Week 24: number analyzed (Participants) | 119 | 123 | 127
  Week 24 | 1.319 (3.0033) | 0.894 (1.5386) | 0.633 (1.0522)

21. Secondary Outcome: ACR Component- Patient's Assessment of Physical Function as Assessed by HAQ-DI Scale Score at Weeks 4, 8, 12, 16, 20 and 24
Description: Patient's assessment of physical function was measured by Disability Index of the Health Assessment Questionnaire (HAQ-DI). HAQ-DI score assess functional status of participant. It is 20 question instrument that assess degree of difficulty a person has in accomplishing tasks in 8 functional areas (dressing, arising, eating, walking, hygiene, reaching, gripping, and activities of daily living). Responses in each functional area were scored from 0=indicating no difficulty, to 3=indicating inability to perform a task in that area. Total HAQ score is average of the computed categories scores ranging from 0-3 where 0=least difficulty and 3=extreme difficulty. Lower scores are indicative of better functioning. Negative change from baseline indicates improvement of physical function.
Time Frame: Weeks 4, 8, 12, 16, 20 and 24
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 126 | 127 | 128
units on a scale
  Week 4: number analyzed (Participants) | 124 | 124 | 128
  Week 4 | 1.2188 (0.67806) | 1.1371 (0.59755) | 0.9824 (0.65278)
  Week 8: number analyzed (Participants) | 123 | 126 | 128
  Week 8 | 1.1331 (0.66928) | 1.0188 (0.61463) | 0.9150 (0.65488)
  Week 12: number analyzed (Participants) | 123 | 126 | 127
  Week 12 | 1.1169 (0.63813) | 0.9831 (0.64058) | 0.8012 (0.63060)
  Week 16: number analyzed (Participants) | 122 | 124 | 127
  Week 16 | 1.1035 (0.65372) | 0.9375 (0.65845) | 0.7776 (0.66011)
  Week 20: number analyzed (Participants) | 118 | 124 | 126
  Week 20 | 1.1049 (0.67838) | 0.8730 (0.62347) | 0.7619 (0.66491)
  Week 24: number analyzed (Participants) | 118 | 123 | 127
  Week 24 | 1.1133 (0.69279) | 0.8770 (0.60691) | 0.7264 (0.63225)

22. Secondary Outcome: Percent Change From Baseline in ACR Components at Weeks 4, 8, 12, 16, 20 and 24
Description: ACR components include swollen joint count (66 joints), tender joint count (68 joints), patient's assessment of pain using visual analog scale (VAS; 0-100 mm, 0=no pain and 100=worst possible pain), patient's global assessment of disease activity (arthritis, VAS; 0-100 mm, 0=excellent and 100= poor), physician's global assessment of disease activity (VAS; 0-100 mm, 0=no arthritis activity and 100=extremely active arthritis), patient's assessment of physical function measured by Disability Index of the Health Assessment Questionnaire (HAQ-DI; a 20-question instrument assessing 8 functional areas; range: 0-3, 0=no difficulty, 3=inability to perform a task in that area), and CRP.
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20 and 24
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 126 | 127 | 128
percent change
  Week 4: Swollen Joint Count: number analyzed (Participants) | 124 | 124 | 128
  Week 4: Swollen Joint Count | -22.4 (49.78) | -27.5 (42.92) | -29.3 (50.85)
  Week 8: Swollen Joint Count: number analyzed (Participants) | 122 | 125 | 128
  Week 8: Swollen Joint Count | -29.4 (50.57) | -45.3 (66.29) | -46.5 (53.81)
  Week 12: Swollen Joint Count: number analyzed (Participants) | 123 | 126 | 127
  Week 12: Swollen Joint Count | -38.1 (55.69) | -60.0 (48.23) | -61.1 (42.62)
  Week 16: Swollen Joint Count: number analyzed (Participants) | 122 | 123 | 127
  Week 16: Swollen Joint Count | -36.6 (56.25) | -65.8 (40.42) | -71.3 (34.69)
  Week 20: Swollen Joint Count: number analyzed (Participants) | 118 | 122 | 126
  Week 20: Swollen Joint Count | -44.4 (54.01) | -66.2 (38.24) | -71.0 (40.88)
  Week 24: Swollen Joint Count: number analyzed (Participants) | 118 | 123 | 127
  Week 24: Swollen Joint Count | -49.5 (45.66) | -66.6 (47.09) | -73.3 (37.95)
  Week 4: Tender Joint Count: number analyzed (Participants) | 124 | 124 | 128
  Week 4: Tender Joint Count | -15.4 (36.11) | -22.2 (36.99) | -17.2 (50.26)
  Week 8: Tender Joint Count: number analyzed (Participants) | 122 | 125 | 128
  Week 8: Tender Joint Count | -21.4 (41.36) | -35.7 (47.45) | -31.4 (47.13)
  Week 12: Tender Joint Count: number analyzed (Participants) | 123 | 126 | 127
  Week 12: Tender Joint Count | -24.5 (50.74) | -48.0 (40.24) | -47.9 (38.76)
  Week 16: Tender Joint Count: number analyzed (Participants) | 122 | 123 | 127
  Week 16: Tender Joint Count | -19.9 (50.84) | -52.6 (36.33) | -49.2 (57.97)
  Week 20: Tender Joint Count: number analyzed (Participants) | 118 | 122 | 126
  Week 20: Tender Joint Count | -30.8 (53.79) | -55.4 (40.17) | -59.4 (35.91)
  Week 24: Tender Joint Count: number analyzed (Participants) | 118 | 123 | 127
  Week 24: Tender Joint Count | -29.1 (53.54) | -53.7 (45.12) | -56.0 (41.76)
  Week 4: Patient's Assessment of Pain: number analyzed (Participants) | 123 | 123 | 127
  Week 4: Patient's Assessment of Pain | 2.98 (38.337) | -2.41 (43.139) | -9.12 (37.068)
  Week 8: Patient's Assessment of Pain: number analyzed (Participants) | 122 | 126 | 127
  Week 8: Patient's Assessment of Pain | -7.41 (42.846) | -12.18 (46.920) | -19.41 (45.862)
  Week 12: Patient's Assessment of Pain: number analyzed (Participants) | 122 | 126 | 126
  Week 12: Patient's Assessment of Pain | -7.82 (49.910) | -22.74 (45.048) | -27.28 (42.305)
  Week 16: Patient's Assessment of Pain: number analyzed (Participants) | 121 | 124 | 126
  Week 16: Patient's Assessment of Pain | -7.86 (47.980) | -25.45 (47.860) | -29.74 (53.817)
  Week 20: Patient's Assessment of Pain: number analyzed (Participants) | 117 | 124 | 125
  Week 20: Patient's Assessment of Pain | -8.31 (54.287) | -29.36 (46.581) | -38.45 (46.235)
  Week 24: Patient's Assessment of Pain: number analyzed (Participants) | 117 | 123 | 126
  Week 24: Patient's Assessment of Pain | -5.35 (53.599) | -32.65 (45.343) | -38.97 (43.873)
  Week 4: PtGA of Disease Activity: number analyzed (Participants) | 124 | 123 | 128
  Week 4: PtGA of Disease Activity | 0.06 (37.022) | -9.57 (30.374) | -2.82 (58.438)
  Week 8: PtGA of Disease Activity: number analyzed (Participants) | 123 | 126 | 128
  Week 8: PtGA of Disease Activity | -9.06 (43.197) | -20.08 (45.707) | -14.95 (46.672)
  Week 12: PtGA of Disease Activity: number analyzed (Participants) | 123 | 126 | 127
  Week 12: PtGA of Disease Activity | -10.00 (49.346) | -28.38 (40.863) | -26.84 (48.800)
  Week 16: PtGA of Disease Activity: number analyzed (Participants) | 122 | 124 | 127
  Week 16: PtGA of Disease Activity | -8.56 (55.279) | -26.93 (42.999) | -30.16 (47.486)
  Week 20: PtGA of Disease Activity: number analyzed (Participants) | 118 | 124 | 126
  Week 20: PtGA of Disease Activity | -11.67 (54.531) | -34.61 (40.905) | -38.76 (43.118)
  Week 24: PtGA of Disease Activity: number analyzed (Participants) | 118 | 123 | 127
  Week 24: PtGA of Disease Activity | -4.91 (65.728) | -37.16 (39.760) | -40.32 (42.037)
  Week 4: PGA of Disease Activity: number analyzed (Participants) | 122 | 123 | 126
  Week 4: PGA of Disease Activity | -10.50 (30.144) | -17.83 (34.370) | -22.42 (34.627)
  Week 8: PGA of Disease Activity: number analyzed (Participants) | 122 | 125 | 128
  Week 8: PGA of Disease Activity | -20.87 (38.908) | -36.57 (34.906) | -41.05 (31.682)
  Week 12: PGA of Disease Activity: number analyzed (Participants) | 122 | 125 | 127
  Week 12: PGA of Disease Activity | -30.47 (32.894) | -40.61 (37.367) | -48.87 (35.082)
  Week 16: PGA of Disease Activity: number analyzed (Participants) | 120 | 123 | 124
  Week 16: PGA of Disease Activity | -29.42 (36.058) | -45.04 (36.363) | -55.36 (32.848)
  Week 20: PGA of Disease Activity: number analyzed (Participants) | 117 | 121 | 125
  Week 20: PGA of Disease Activity | -36.48 (35.490) | -51.88 (34.491) | -59.57 (30.353)
  Week 24: PGA of Disease Activity: number analyzed (Participants) | 117 | 122 | 127
  Week 24: PGA of Disease Activity | -33.95 (34.349) | -53.43 (37.305) | -61.39 (31.234)
  Week 4: HAQ-DI Score: number analyzed (Participants) | 118 | 121 | 119
  Week 4: HAQ-DI Score | 4.3521 (61.86548) | -0.4964 (54.63888) | -5.9245 (53.44204)
  Week 8: HAQ-DI Score: number analyzed (Participants) | 117 | 123 | 119
  Week 8: HAQ-DI Score | -3.3329 (48.15101) | -9.1556 (65.76295) | -11.3467 (69.07565)
  Week 12: HAQ-DI Score: number analyzed (Participants) | 117 | 123 | 118
  Week 12: HAQ-DI Score | -2.1600 (88.42239) | -13.1115 (69.57297) | -21.6242 (65.32053)
  Week 16: HAQ-DI Score: number analyzed (Participants) | 116 | 122 | 118
  Week 16: HAQ-DI Score | -3.2447 (109.78825) | -19.5421 (55.80512) | -27.7444 (68.28273)
  Week 20: HAQ-DI Score: number analyzed (Participants) | 112 | 122 | 118
  Week 20: HAQ-DI Score | -10.5259 (44.67386) | -23.6139 (65.27566) | -26.2478 (74.38446)
  Week 24: HAQ-DI Score: number analyzed (Participants) | 112 | 121 | 118
  Week 24: HAQ-DI Score | -7.3745 (61.62081) | -8.7950 (148.19861) | -31.1750 (72.70079)
  Week 4: CRP: number analyzed (Participants) | 124 | 123 | 128
  Week 4: CRP | 9.972 (66.9599) | -4.060 (76.1801) | -1.054 (102.5692)
  :Week 8: CRP: number analyzed (Participants) | 120 | 124 | 127
  :Week 8: CRP | 10.402 (83.4766) | 5.403 (111.6889) | 11.791 (273.1510)
  Week 12: CRP: number analyzed (Participants) | 122 | 123 | 127
  Week 12: CRP | 9.295 (94.9020) | -2.507 (98.4549) | -7.908 (114.4983)
  Week 16: CRP: number analyzed (Participants) | 120 | 123 | 124
  Week 16: CRP | 82.057 (734.6577) | 7.139 (134.6682) | 2.759 (208.7305)
  Week 20: CRP: number analyzed (Participants) | 119 | 124 | 126
  Week 20: CRP | 5.768 (98.6914) | -11.151 (84.9807) | -14.684 (98.0041)
  Week 24: CRP: number analyzed (Participants) | 119 | 123 | 127
  Week 24: CRP | 31.628 (239.7722) | -7.404 (101.4807) | -6.112 (148.2088)

23. Secondary Outcome: Change From Baseline in HAQ-DI Score at Weeks 4, 8, 12, 16, 20 and 24
Description: as for outcome 2
Time Frame: Baseline, Week 4, 8, 12, 16, 20 and 24
Population: as for outcome 6
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 126 | 127 | 128
units on a scale
  Week 4 | 0.0043 [-0.0562 to 0.0647] | -0.0571 [-0.1173 to 0.0031] | -0.1095 [-0.1695 to -0.0494]
  Week 8 | -0.0781 [-0.1498 to -0.0064] | -0.1711 [-0.2423 to -0.0999] | -0.1907 [-0.2619 to -0.1194]
  Week 12 | -0.1013 [-0.1783 to -0.0243] | -0.2174 [-0.2938 to -0.1410] | -0.3209 [-0.3973 to -0.2444]
  Week 16 | -0.1131 [-0.1955 to -0.0307] | -0.2620 [-0.3438 to -0.1802] | -0.3393 [-0.4211 to -0.2575]
  Week 20 | -0.1079 [-0.1935 to -0.0223] | -0.3293 [-0.4143 to -0.2443] | -0.3708 [-0.4558 to -0.2858]
  Week 24 | -0.0743 [-0.1605 to -0.0119] | -0.3225 [-0.4082 to -0.2369] | -0.3968 [-0.4825 to -0.3112]

24. Secondary Outcome: Percentage of Participants Who Achieved a Clinically Meaningful Improvement (>=0.35 Improvement From Baseline) in HAQ-DI Score by Visit Over Time Through Week 24 Among Participants With HAQ-DI Score >=0.35 at Baseline
Description: HAQ-DI score assess functional status of participant. It is 20 question instrument that assess degree of difficulty a person has in accomplishing tasks in 8 functional areas (dressing, arising, eating, walking, hygiene, reaching, gripping, and activities of daily living). Responses in each functional area were scored from 0=indicating no difficulty, to 3=indicating inability to perform a task in that area. Total HAQ score is average of the computed categories scores ranging from 0-3, where 0=least difficulty and 3=extreme difficulty. Lower scores are indicative of better functioning. Negative change from baseline indicates improvement of physical function and a decrease of 0.35 from baseline in HAQ-DI score indicates a meaningful improvement.
Time Frame: Week 4, 8, 12, 16, 20 and 24
Population: FAS1 among the participants with HAQ-DI Score >=0.35 at baseline. Participants with HAQ-DI >=0.35 improvement from baseline at specific timepoint and did not meet any TF criteria before, considered responders at that time point. Participants who met 1 or more TF criteria before or with missing data at that time point were considered non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 110 | 112 | 110
percentage of participants
  Week 4 | 20.0 | 26.8 | 30.9
  Week 8 | 25.5 | 40.2 | 38.2
  Week 12 | 27.3 | 45.5 | 51.8
  Week 16 | 30.9 | 46.4 | 57.3
  Week 20 | 28.2 | 50.9 | 56.4
  Week 24 | 29.1 | 50.9 | 57.3

25. Secondary Outcome: Percentage of Participants Who Achieved a DAS28 (CRP) Response by Visit Over Time Through Week 24
Description: DAS28 based on CRP is an index combining tender joints (28 joints), swollen joints (28 joints), CRP and patient's global assessment of disease activity. The set of 28 joint count is based on evaluation of the shoulder, elbow, wrist, metacarpophalangeal (MCP) MCP1 to MCP5, proximal interphalangeal (PIP) PIP1 to PIP5 joints of both the upper right extremity and the upper left extremity as well as the knee joints of lower right and lower left extremities. DAS28 (CRP) response criteria was defined as follows: Good response: less than or equal to (<=) 3.2 at visit and >1.2 improvement; Moderate response: >3.2 at visit and >1.2 improvement or <=5.1 at visit and >0.6-1.2 improvement; No response: <=0.6 improvement, or >5.1 at visit and <=1.2 improvement. The values are 0=best to 10=worst. A DAS28 (CRP) responder was defined as achieving a good or moderate DAS28 response at a specific visit.
Time Frame: Weeks 4, 8, 12, 16, 20 and 24
Population: Analysis population is FAS1. Participants who achieved DAS28 (CRP) response at a specific timepoint and did not meet any TF criteria before, were considered as responders at that time point. Participants who met 1 or more TF criteria before or with missing data at that time point were considered as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 126 | 127 | 128
percentage of participants
  Week 4 | 27.0 | 33.1 | 40.6
  Week 8 | 35.7 | 59.1 | 54.7
  Week 12 | 41.3 | 67.7 | 74.2
  Week 16 | 44.4 | 65.4 | 73.4
  Week 20 | 46.0 | 66.1 | 75.0
  Week 24 | 44.4 | 70.9 | 76.6

26. Secondary Outcome: Percentage of Participants Who Achieved a DAS28 (CRP) Remission by Visit Over Time Through Week 24
Description: DAS28 based on CRP is an index combining tender joints (28 joints), swollen joints (28 joints), CRP and patient's global assessment of disease activity. The set of 28 joint count is based on evaluation of the shoulder, elbow, wrist, metacarpophalangeal (MCP) MCP1 to MCP5, proximal interphalangeal (PIP) PIP1 to PIP5 joints of both the upper right extremity and the upper left extremity as well as the knee joints of lower right and lower left extremities. The values are 0=best to 10=worst. DAS 28 (CRP) remission was defined as DAS 28 (CRP) value <2.6 at the analysis visit.
Time Frame: Week 4, 8, 12, 16, 20 and 24
Population: Analysis population is FAS1. Participants who achieved DAS28 (CRP) remission at a specific timepoint and did not meet any TF criteria before, were considered as responders at that time point. Participants who met 1 or more TF criteria before or with missing data at that time point were considered as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 126 | 127 | 128
percentage of participants
  Week 4 | 3.2 | 7.9 | 7.8
  Week 8 | 7.9 | 11.0 | 11.7
  Week 12 | 9.5 | 22.0 | 21.9
  Week 16 | 7.9 | 19.7 | 25.0
  Week 20 | 17.5 | 25.2 | 36.7
  Week 24 | 12.7 | 23.6 | 35.9

27. Secondary Outcome: Change From Baseline in DAS28 (CRP) Score at Weeks 4, 8, 12, 16, 20 and 24
Description: DAS28 based on CRP is an index combining tender joints (28 joints), swollen joints (28 joints), CRP and patient's global assessment of disease activity. The set of 28 joint count is based on evaluation of the shoulder, elbow, wrist, metacarpophalangeal (MCP) MCP1 to MCP5, proximal interphalangeal (PIP) PIP1 to PIP5 joints of both the upper right extremity and the upper left extremity as well as the knee joints of lower right and lower left extremities. The values are 0=best to 10=worst. Negative change from baseline indicates improvement of arthritis.
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20 and 24
Population: as for outcome 6
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 126 | 127 | 128
units on a scale
  Week 4 | -0.35 [-0.48 to -0.22] | -0.53 [-0.67 to -0.40] | -0.56 [-0.69 to -0.43]
  Week 8 | -0.55 [-0.71 to -0.39] | -0.83 [-0.99 to -0.67] | -0.88 [-1.04 to -0.72]
  Week 12 | -0.63 [-0.80 to -0.47] | -1.16 [-1.33 to -0.99] | -1.23 [-1.39 to -1.06]
  Week 16 | -0.64 [-0.82 to -0.46] | -1.19 [-1.37 to -1.01] | -1.38 [-1.56 to -1.20]
  Week 20 | -0.80 [-1.00 to -0.60] | -1.38 [-1.58 to -1.19] | -1.56 [-1.76 to -1.37]
  Week 24 | -0.70 [-0.89 to -0.51] | -1.43 [-1.61 to -1.24] | -1.61 [-1.80 to -1.42]

28. Secondary Outcome: Percentage of Participants Who Achieved a Response Based on Modified Psoriatic Arthritis Responder Criteria (PsARC) by Visit Over Time Through Week 24
Description: The modified PsARC response was defined as improvement in at least 2 of the four criteria: >=30% decrease in swollen joint count, >=30% decrease in tender joint count, >=20% improvement in patient's Global Assessment of Disease Activity (arthritis) using VAS (0-100 mm, 0=excellent and 100= poor), >=20% improvement in physician's Global Assessment of Disease Activity using VAS (VAS: 0-100 mm, 0=no arthritis activity and 100=extremely active arthritis), and at least one of the 2 joint criteria with no deterioration in the other criteria.
Time Frame: Weeks 4, 8, 12, 16, 20 and 24
Population: Analysis population is FAS1. Participants who achieved a modified PsARC response at a specific time point and did not meet any TF criteria before, were considered as responders at that time point. Participants who met 1 or more TF criteria before or with missing data at that time point were considered as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 126 | 127 | 128
percentage of participants
  Week 4 | 20.6 | 29.1 | 33.6
  Week 8 | 32.5 | 56.7 | 48.4
  Week 12 | 41.3 | 58.3 | 66.4
  Week 16 | 36.5 | 64.6 | 68.0
  Week 20 | 41.3 | 66.1 | 75.8
  Week 24 | 31.0 | 59.8 | 72.7

29. Secondary Outcome: Percentage of Participants Who Achieved Resolution of Enthesitis at Weeks 4, 8, 16, and 24 Among the Participants With Enthesitis at Baseline
Description: Enthesitis was assessed using the LEI, a tool developed to assess enthesitis in participants with PsA and evaluates the presence (score of 1) or absence (score of 0) of pain by applying local pressure to the following entheses: left and right lateral epicondyle humerus, left and right medial femoral condyle, and left and right achilles tendon insertion. The enthesitis index score is a total score of the 6 evaluated sites from 0 (0 sites with tenderness) to 6 (worst possible score; 6 sites with tenderness). A LEI score of 0 at a post baseline visit indicates resolution of enthesitis when baseline LEI>0.
Time Frame: Weeks 4, 8, 16, and 24
Population: FAS1 among the participants with enthesitis at baseline. Participants who achieved enthesitis resolution at a specific timepoint and did not meet any TF criteria before, were considered as responders at that time point. Participants who met 1 or more TF criteria before or with missing data at that time point were considered as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 77 | 72 | 73
percentage of participants
  Week 4 | 22.1 | 18.1 | 27.4
  Week 8 | 23.4 | 30.6 | 30.1
  Week 16 | 37.7 | 34.7 | 45.2
  Week 24 | 27.3 | 40.3 | 47.9

30. Secondary Outcome: Change From Baseline in Enthesitis Score at Weeks 4, 8, 16 and 24 Among the Participants With Enthesitis at Baseline
Description: Enthesitis was assessed using the LEI, a tool developed to assess enthesitis in participants with PsA and evaluates the presence (score of 1) or absence (score of 0) of pain by applying local pressure to the following entheses: left and right lateral epicondyle humerus, left and right medial femoral condyle, and left and right achilles tendon insertion. The enthesitis index score is a total score of the 6 evaluated sites from 0 (0 sites with tenderness) to 6 (worst possible score; 6 sites with tenderness). Negative changes from baseline indicate improvement of enthesitis.
Time Frame: Baseline, Weeks 4, 8, 16 and 24
Population: Analysis population is FAS1 among the participants with enthesitis at baseline. Data after meeting one or more TF criteria were imputed as no change from baseline. Missing data were assumed to be MAR and imputed using MI.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 77 | 72 | 73
units on a scale
  Week 4 | -0.37 [-0.69 to -0.05] | -0.45 [-0.78 to -0.11] | -0.96 [-1.30 to -0.62]
  Week 8 | -0.65 [-1.00 to -0.31] | -0.83 [-1.19 to -0.47] | -1.11 [-1.48 to -0.74]
  Week 16 | -0.99 [-1.36 to -0.61] | -1.00 [-1.39 to -0.61] | -1.51 [-1.90 to -1.11]
  Week 24 | -1.01 [-1.37 to -0.66] | -1.35 [-1.72 to -0.98] | -1.75 [-2.13 to -1.38]

31. Secondary Outcome: Percentage of Participants With Resolution of Dactylitis by Visit Over Time Through Week 24 Among the Participants With Dactylitis at Baseline
Description: as for outcome 13
Time Frame: Weeks 4, 8, 16 and 24
Population: FAS1 among the participants with dactylitis at baseline. Participants who achieved dactylitis resolution at a specific timepoint and did not meet any TF criteria before, were considered as responders at that time point. Participants who met 1 or more TF criteria before or with missing data at that time point were considered as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 55 | 49 | 38
percentage of participants
  Week 4 | 41.8 | 34.7 | 31.6
  Week 8 | 41.8 | 40.8 | 44.7
  Week 16 | 43.6 | 59.2 | 57.9
  Week 24 | 49.1 | 65.3 | 63.2

32. Secondary Outcome: Change From Baseline in Dactylitis Score at Weeks 4, 8, 16 and 24 Among the Participants With Dactylitis at Baseline
Description: The presence and severity of dactylitis was assessed in both hands and feet using a scoring system from 0 to 3 (0-no dactylitis, 1-mild dactylitis, 2-moderate dactylitis, and 3-severe dactylitis) for each digit. The results were summed to produce a final score ranging from 0 to 60. A higher score indicates more severe dactylitis. Negative changes from baseline indicate improvement in dactylitis.
Time Frame: Baseline, Weeks 4, 8, 16 and 24
Population: as for outcome 14
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 55 | 49 | 38
units on a scale
  Week 4 | -2.77 [-4.24 to -1.30] | -2.24 [-3.76 to -0.72] | -2.63 [-4.39 to -0.86]
  Week 8 | -2.92 [-4.58 to -1.26] | -4.00 [-5.72 to -2.29] | -3.92 [-5.90 to -1.93]
  Week 16 | -4.03 [-5.76 to -2.30] | -6.00 [-7.79 to -4.22] | -6.29 [-8.36 to -4.22]
  Week 24 | -4.30 [-5.96 to -2.63] | -6.11 [-7.81 to -4.41] | -5.82 [-7.82 to -3.83]

33. Secondary Outcome: Change From Baseline in the Psoriatic Arthritis Disease Activity (PASDAS) Score at Weeks 8, 16 and 24
Description: PASDAS (score range of 0 to 10, where higher score indicated more severe disease) is a compositive score of overall disease activity combining Patient's Global Assessment of Disease Activity (arthritis and psoriasis, using VAS [0-100 mm, 0=excellent and 100= poor), Physician's Global Assessment of Disease Activity (using VAS [0-100 mm, 0=no arthritis activity and 100=extremely active arthritis]), swollen joint count (0-66 joints), tender joint count (0-68 joints), CRP (mg/L), enthesitis based on LEI (0-6), tender dactylitis count (scoring each digit from 0-3 and recoding to 0-1, where any score > 0 equaled 1), and the PCS score of the SF-36 health survey. The cutoffs for disease activity were 3.2 (low) to 5.4 (high). Negative changes from baseline indicate improvement of overall disease activity.
Time Frame: Baseline, Weeks 8, 16 and 24
Population: Analysis population is FAS1. Data after meeting one or more TF criteria were imputed as no change from baseline. Missing data were assumed to be MAR. The LS mean is based on Mixed-effect repeated measures (MMRM) model that included data from all visits for all participants included in the model.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 126 | 127 | 128
units on a scale
  Week 8 | -0.759 [-0.961 to -0.556] | -1.315 [-1.518 to -1.113] | -1.428 [-1.628 to -1.228]
  Week 16 | -0.980 [-1.221 to -0.739] | -1.779 [-2.019 to -1.539] | -2.083 [-2.322 to -1.843]
  Week 24 | -0.959 [-1.212 to -0.707] | -2.124 [-2.376 to -1.871] | -2.407 [-2.657 to -2.156]

34. Secondary Outcome: Change From Baseline in Group of Research and Assessment of Psoriasis and Psoriatic Arthritis Composite (GRACE) Score at Weeks 16 and 24
Description: GRACE index is a composite PsA disease activity score converted from Arithmetic Mean of Desirability Function (AMDF), derived from TJC (0-68) and SJC (0-66), HAQ-DI (0-3), patient's global assessment of disease activity on arthritis and psoriasis (0-100 mm, 0=excellent and 100=poor), patient's assessment of skin disease activity (0-100 mm, 0=excellent and 100=poor), patient's global assessment of disease activity on arthritis (0-100 mm, 0=excellent and 100=poor), PASI (0-72), and PsA Quality of Life Index (derived as PsAQOL=25.355 + [2.367*HAQ-DI]-[0.234*SF-PCS]-[0.244*SF-MCS]), where HAQ-DI: HAQ-DI score (0-3, 0=least difficulty and 3=extreme difficulty), SF-PCS (Score ranges from 0-100, higher scores= better quality of life) and SF-MCS (score ranges from 0-100, higher scores= better quality of life). Total score is from 0-10, lower score=better response. Higher score indicates more active disease activity. Negative change from baseline indicates improvement of PsA disease activity.
Time Frame: Baseline, Weeks 16 and 24
Population: Analysis population is FAS1. Data after meeting one or more TF criteria were imputed as no change from baseline. Missing data were assumed to be MAR. LS mean is based on MMRM model that included data from all visits for all participants included in model. Here, n (number analyzed) signifies number of participants analyzed at specified timepoints.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 126 | 127 | 128
units on a scale
  Week 16 | -0.918 [-1.176 to -0.659] | -2.024 [-2.283 to -1.765] | -2.368 [-2.625 to -2.111]
  Week 24 | -0.854 [-1.122 to -0.586] | -2.368 [-2.636 to -2.099] | -2.735 [-3.001 to -2.468]

35. Secondary Outcome: Change From Baseline in the Disease Activity Index for Psoriatic Arthritis (DAPSA) Score at Weeks 4, 8, 12, 16, 20 and 24
Description: DAPSA assessed the joint domain of psoriatic arthritis (PsA) and was derived from the sum of the following components: tender joint count (0-68), swollen joint count (0-66), CRP level (mg/dL, value <lower limit of quantification [LLOQ] is considered equal to half of the value of LLOQ for numerical calculations), patient assessment of pain (0-10 centimeter [cm] VAS, 0=no pain, 10=worst possible pain), and patient's global assessment of disease activity on arthritis (0 to 10 cm VAS, 0=excellent and 10=poor). A higher score indicates more active disease activity. Negative changes from baseline indicate improvement of PsA disease activity. The assessment does not have a score range with an upper or lower bound.
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20 and 24
Population: Analysis population is FAS1. Data after meeting one or more TF criteria were imputed as no change from baseline. Missing data were assumed to be MAR. The LS mean is based on MMRM model that included data from all visits for all participants included in the model.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 126 | 127 | 128
units on a scale
  Week 4 | -4.826 [-6.901 to -2.752] | -7.815 [-9.926 to -5.705] | -8.574 [-10.636 to -6.511]
  Week 8 | -8.776 [-11.307 to -6.246] | -13.601 [-16.118 to -11.084] | -13.231 [-15.731 to -10.732]
  Week 12 | -10.135 [-12.670 to -7.599] | -18.167 [-20.704 to -15.631] | -17.433 [-19.949 to -14.918]
  Week 16 | -9.964 [-12.568 to -7.359] | -19.830 [-22.426 to -17.234] | -19.389 [-21.977 to -16.802]
  Week 20 | -11.552 [-14.228 to -8.876] | -20.570 [-23.248 to -17.891] | -21.244 [-23.903 to -18.586]
  Week 24 | -10.749 [-13.396 to -8.102] | -21.332 [-23.977 to -18.688] | -20.621 [-23.251 to -17.992]

36. Secondary Outcome: Percentage of Participants Who Achieved Minimal Disease Activity (MDA) at Weeks 16 and 24
Description: MDA was considered achieved if at least 5 of the following 7 criteria were met at the analysis visit: tender joint count <=1; swollen joint count <=1; psoriasis activity and severity index <=1; patient's assessment of pain VAS score of <=15; patient's global assessment of disease activity VAS (arthritis and psoriasis) score of <=20; HAQ-DI <=0.5; and tender entheseal points <=1.
Time Frame: Weeks 16 and Week 24
Population: Analysis population is FAS1. Participants who achieved MDA at a specific timepoint and did not meet any TF criteria before, were considered as responders at that time point. Participants who met 1 or more TF criteria before or with missing data at that time point were considered as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 126 | 127 | 128
percentage of participants
  Week 16 | 7.1 | 15.7 | 18.0
  Week 24 | 11.1 | 22.8 | 30.5

37. Secondary Outcome: Percentage of Participants Who Achieved >= 20%, >=50%, >=70%, and >=90% Improvement From Baseline in BASDAI Score Through Week 24 Among the Participants With Spondylitis and Peripheral Arthritis and BASDAI Score >0 at Baseline
Description: Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) is a self-assessment tool that consists of 6 questions relating to the 5 major symptoms of ankylosing spondylitis: fatigue, spinal pain, joint pain, enthesitis, qualitative morning stiffness and quantitative morning stiffness. The first 5 items were scored on a 10 centimeter (cm) VAS ranging from 0=none to 10=very severe. Quantitative morning stiffness was scored on a 10cm VAS ranging from 0=0 hours to 10=2 or more hours. The 2 scores for qualitative and quantitative morning stiffness were averaged, and the total BASDAI score was the average of the 5 scores of each symptom, ranging from 0 (none) to 10 (very severe). Higher scores indicate greater disease severity and an improvement of 50% from baseline is considered clinically meaningful. Only participants with spondylitis with peripheral arthritis as their primary arthritic presentation of PsA completed the BASDAI indicate the degree of their symptoms over the past week.
Time Frame: Weeks 8, 16 and 24
Population: FAS1 with spondylitis and peripheral arthritis and BASDAI score >0 at baseline. Participants with the specified improvement in BASDAI at specific time point and did not meet TF criteria before, considered responders at that time point. Participants who met 1/more TF criteria before or with missing data at that time point considered non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 23 | 24 | 20
percentage of participants
  Week 8: Participants with >=20% Improvement | 26.1 | 58.3 | 55.0
  Week 16: Participants with >=20% Improvement | 52.2 | 75.0 | 65.0
  Week 24: Participants with >=20% Improvement | 26.1 | 70.8 | 65.0
  Week 8: Participants with >=50% Improvement | 4.3 | 25.0 | 25.0
  Week 16: Participants with >=50% Improvement | 26.1 | 29.2 | 35.0
  Week 24: Participants with >=50% Improvement | 13.0 | 41.7 | 35.0
  Week 8: Participants with >=70% Improvement | 4.3 | 4.2 | 15.0
  Week 16: Participants with >=70% Improvement | 8.7 | 25.0 | 15.0
  Week 24: Participants with >=70% Improvement | 8.7 | 29.2 | 5.0
  Week 8: Participants with >=90% Improvement | 0 | 0 | 0
  Week 16: Participants with >=90% Improvement | 0 | 8.3 | 10.0
  Week 24: Participants with >=90% Improvement | 0 | 16.7 | 0

38. Secondary Outcome: Change From Baseline in BASDAI Score at Week 8, 16, and Week 24 Among Participants With Spondylitis and Peripheral Arthritis at Baseline
Description: as for outcome 37
Time Frame: Baseline, Weeks 8, 16, and 24
Population: Analysis population is FAS1 among the participants with spondylitis and peripheral arthritis at baseline. Data after meeting one or more TF criteria were imputed as no change from baseline. Missing data were assumed to be MAR. The LS mean is based on MMRM model that included data from all visits for all participants included in the model.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 23 | 24 | 20
units on a scale
  Week 8 | -0.595 [-1.351 to -0.162] | -1.577 [-2.296 to -0.859] | -1.976 [-2.779 to -1.174]
  Week 16 | -1.604 [-2.483 to -0.725] | -2.419 [-3.261 to -1.577] | -2.469 [-3.405 to -1.533]
  Week 24 | -0.919 [-1.795 to -0.043] | -2.665 [-3.503 to -1.826] | -2.074 [-3.006 to -1.142]

39. Secondary Outcome: Percentage of Participants With Low or Very Low Disease Activity Based on Psoriatic Arthritis Disease Activity Score (PASDAS) by Visit Over Time Through Week 24
Description: PASDAS (score range of 0 to 10, where higher score indicated more severe disease) is a compositive score of overall disease activity combining Patient's Global Assessment of Disease Activity (arthritis and psoriasis, using VAS [0-100 mm, 0=excellent and 100= poor), Physician's Global Assessment of Disease Activity (using VAS [0-100 mm, 0=no arthritis activity and 100=extremely active arthritis]), swollen joint count (0-66 joints), tender joint count (0-68 joints), CRP (mg/L), enthesitis based on LEI (0-6), tender dactylitis count (scoring each digit from 0-3 and recoding to 0-1, where any score > 0 equaled 1), and the PCS score of the SF-36 health survey. The cutoffs for disease activity were 3.2 (low) to 5.4 (high).
Time Frame: Weeks 8, 16 and 24
Population: Analysis population is FAS1. Participants with low or very low disease activity at a specific timepoint and did not meet any TF criteria before, were considered as responders at that time point. Participants who met 1 or more TF criteria before or with missing data at that time point were considered as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 126 | 127 | 128
percentage of participants
  Week 8 | 4.0 | 10.2 | 14.8
  Week 16 | 8.7 | 22.0 | 27.3
  Week 24 | 11.1 | 30.7 | 36.7

40. Secondary Outcome: Percentage of Participants With Low Disease Activity Based on Group of Research and Assessment of Psoriasis and Psoriatic Arthritis Composite (GRACE) Score Index by Visit Over Time Through Week 24
Description: GRACE index is a composite PsA disease activity score converted from Arithmetic Mean of the Desirability Function (AMDF), which was derived from TJC (0-68) and SJC (0-66), HAQ-DI (0-3), patient's global assessment of disease activity on arthritis and psoriasis (0-100 mm, 0=excellent and 100= poor), patient's assessment of skin disease activity (0-100 mm, 0=excellent and 100=poor), patient's global assessment of disease activity on arthritis (0-100 mm, 0=excellent and 100=poor), PASI (0-72), and PsA Quality of Life Index (derived as PsAQOL =25.355 + [2.367*HAQ-DI] - [0.234*SF-PCS] - [0.244*SF-MCS]), where HAQ-DI: HAQ-DI score (0-3, 0=least difficulty and 3=extreme difficulty), SF-PCS (Score ranges from 0 to 100, higher scores= better quality of life) and SF-MCS (score ranges from 0 to 100, higher scores= better quality of life). The total score is from 0-10, where lower score indicates better response. Higher score indicates more active disease activity.
Time Frame: Weeks 16 and 24
Population: Analysis population is FAS1. Participants with low disease activity at a specific timepoint and did not meet any TF criteria before, were considered as responders at that time point. Participants who met 1 or more TF criteria before or with missing data at that time point were considered as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 126 | 127 | 128
percentage of participants
  Week 16 | 10.3 | 22.0 | 28.9
  Week 24 | 11.9 | 30.7 | 42.2

41. Secondary Outcome: Percentage of Participants With Low Disease Activity or Remission Based on Disease Activity Index for Psoriatic Arthritis (DAPSA) by Visit Over Time Through Week 24
Description: DAPSA assessed the joint domain of PsA and was derived from the sum of the following components: tender joint count (0-68), swollen joint count (0-66), CRP level (mg/dL), patient assessment of pain (0-10 cm VAS, 0=no pain, 10=worst possible pain), and patient's global assessment of disease activity on arthritis (0 to 10 cm VAS, 0=excellent and 10=poor). A higher score indicates more active disease activity. The assessment does not have a score range with an upper or lower bound.
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20 and 24
Population: Analysis population is FAS1. Participants with low disease activity or remission at a specific timepoint and did not meet any TF criteria before, were considered as responders at that time point. Participants who met 1 or more TF criteria before or with missing data at that time point were considered as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 126 | 127 | 128
percentage of participants
  Baseline | 1.6 | 2.4 | 0.8
  Week 4 | 10.3 | 8.7 | 13.3
  Week 8 | 13.5 | 17.3 | 25.0
  Week 12 | 18.3 | 27.6 | 37.5
  Week 16 | 13.5 | 29.9 | 36.7
  Week 20 | 22.2 | 37.8 | 46.1
  Week 24 | 16.7 | 40.9 | 49.2

42. Secondary Outcome: Percentage of Participants With Very Low Disease Activity (VLDA) by Visit Over Time Through Week 24
Description: A measurement that defines a satisfactory state of disease activity that includes the 5 domains of PsA (joint symptoms, skin psoriasis, patient's perspective of pain and disease activity, physical function, and enthesitis). A participant was considered as having achieved VLDA at a visit if the participant fulfilled all 7 criteria (tender joint count <=1; swollen joint count <=1; PASI <=1; patient pain VAS score of <=15; patient global disease activity VAS [arthritis and psoriasis] score of <=20; Health Assessment Questionnaire (HAQ) score <=0.5; and tender entheseal points <=1) at that visit.
Time Frame: Weeks 16 and 24
Population: Analysis population is FAS1. Participants who achieved VLDA response at a specific timepoint and did not meet any TF criteria before, were considered as responders at that time point. Participants who met 1 or more TF criteria before or with missing data at that time point were considered as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 126 | 127 | 128
percentage of participants
  Week 16 | 2.4 | 3.1 | 3.1
  Week 24 | 1.6 | 3.9 | 9.4

43. Secondary Outcome: Percentage of Participants Who Achieved PASI 75 Response at Weeks 16 and 24 Among Participants With >=3% BSA Psoriatic Involvement and an IGA Score of >=2 at Baseline
Description: PASI is a tool to assess and grade severity of psoriasis and response to therapy. In PASI, body is divided into 4 areas: head, trunk, upper extremities, lower extremities. Each area was assessed separately for percentage of area involved and translated to numeric score ranging from 0 (no involvement) to 6 (90 to 100% involvement), and for erythema, induration, and scaling, each rated on scale of 0 to 4 that is none to maximum severtiy. PASI numeric score range from 0 (no psoriasis) to 72. Higher scores indicate more severe disease. A PASI 75 response: >=75% improvement in PASI score from baseline.
Time Frame: Weeks 16 and 24
Population: FAS1 among participants with >=3% BSA of psoriasis and IGA score >=2 at baseline. Participants with PASI 75 response at specific time point and did not meet any TF criteria before, were considered responders at that time point. Participants who met 1/more TF criteria before or with missing data at that time point were considered non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 78 | 82 | 89
percentage of participants
  Week 16 | 20.5 | 63.4 | 73.0
  Week 24 | 14.1 | 75.6 | 86.5

44. Secondary Outcome: Percentage of Participants Who Achieved PASI 90 Response at Weeks 16 and 24 Among Participants With >=3% BSA Psoriatic Involvement and an IGA Score of >=2 at Baseline
Description: PASI is a tool to assess and grade severity of psoriasis and response to therapy. In PASI, body is divided into 4 areas: head, trunk, upper extremities, lower extremities. Each area was assessed separately for percentage of area involved and translated to numeric score ranging from 0 (no involvement) to 6 (90 to 100% involvement), and for erythema, induration, and scaling, each rated on scale of 0 to 4 that is none to maximum severtiy. PASI numeric score range from 0 (no psoriasis) to 72. Higher scores indicate more severe disease. A PASI 90 response: >=90% improvement in PASI score from baseline.
Time Frame: Weeks 16 and 24
Population: FAS1 among participants with >=3% BSA of psoriasis and IGA score >=2 at baseline. Participants with PASI 90 response at specific time point and did not meet any TF criteria before, were considered responders at that time point. Participants who met 1 or more TF criteria before or with missing data at that time point were considered non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 78 | 82 | 89
percentage of participants
  Week 16 | 10.3 | 45.1 | 52.8
  Week 24 | 11.5 | 50.0 | 62.9

45. Secondary Outcome: Percentage of Participants Who Achieved PASI 100 Response by Visit Over Time Through Week 24 Among Participants With >=3% BSA Psoriatic Involvement and an IGA Score of >=2 at Baseline
Description: PASI is a tool to assess and grade severity of psoriasis and response to therapy. In PASI, body is divided into 4 areas: head, trunk, upper extremities, lower extremities. Each area was assessed separately for percentage of area involved and translated to numeric score ranging from 0 (no involvement) to 6 (90 to 100% involvement), and for erythema, induration, and scaling, each rated on scale of 0 to 4 that is none to maximum severtiy. PASI numeric score range from 0 (no psoriasis) to 72. Higher scores indicate more severe disease. A PASI 100 response: 100% improvement in PASI score from baseline.
Time Frame: Weeks 16 and 24
Population: FAS1 among participants with >=3% BSA of psoriasis and IGA score >=2 at baseline. Participants with PASI 100 response at specific time point and did not meet any TF criteria before, were considered responders at that time point. Participants who met 1/more TF criteria before or with missing data at that time point were considered non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 78 | 82 | 89
percentage of participants
  Week 16 | 7.7 | 23.2 | 32.6
  Week 24 | 6.4 | 25.6 | 44.9

46. Secondary Outcome: Percentage of Participants Who Achieved Both PASI 75 and ACR 20 Responses at Weeks 16 and 24 Among the Participants With >=3% BSA Psoriatic Involvement and an IGA Score of >=2 (Mild) at Baseline
Description: In PASI, each area (head, trunk, upper and lower extremities) was assessed for % of area involved and translated to numeric score from 0 (no involvement) to 6 (90-100% involvement) and for erythema, induration, and scaling, each rated on scale of 0 to 4 that is none to maximum severtiy. PASI produces numeric score from 0 to 72. Higher scores=more severe disease. PASI 75: >=75% improvement in PASI score from baseline. ACR 20: >=20% improvement in swollen joint count (SJC) (66 joints) + tender joint count (TJC) (68 joints) and >=20% improvement in 3 of 5: patient's assessment of pain (VAS; 0-100 mm, 0=no pain to 100=worst possible pain), PtGA of disease activity (VAS; 0-100 mm, 0=excellent to 100=poor), PGA of disease activity (VAS; 0-100 mm, 0=no arthritis to 100=extremely active arthritis), patient's assessment of physical function (HAQ-DI -20-question instrument; range- 0=no difficulty to 3=inability to perform task) and CRP.
Time Frame: Weeks 16 and 24
Population: FAS1 participants with >=3% BSA psoriatic involvement and IGA score >=2 at baseline. Participants with both PASI75 and ACR20 responses at specific timepoint and did not meet TF criteria before, considered responders at that time point. Participants who met 1/more TF criteria before or with missing data at that time point considered non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 78 | 82 | 89
percentage of participants
  Week 16 | 6.4 | 35.4 | 48.3
  Week 24 | 6.4 | 40.2 | 52.8

47. Secondary Outcome: Percentage of Participants Who Achieved Both PASI 75 and Modified PsARC Response by Visit Over Time Through Week 24 Among Participants With >=3% BSA Psoriatic Involvement and an IGA Score of >=2 (Mild) at Baseline
Description: In PASI, each area (head, trunk, upper and lower extremities) was assessed separately for % of area involved and translated to numeric score ranging from 0 (no involvement) to 6 (90-100% involvement), and for erythema, induration, and scaling, each rated on scale of 0 to 4 that is none to maximum severtiy. PASI produces numeric score range from 0 to 72. Higher scores=more severe disease. PASI 75 response: >=75% improvement in PASI score from baseline. Modified PsARC response: improvement in at least 2 of 4 criteria: >=30% decrease in SJC and TJC, >=20% improvement in PtGA of Disease Activity (arthritis) on VAS (0-100 mm, 0=excellent and 100=poor), >=20% improvement in PGA of Disease Activity on VAS (VAS: 0-100 mm, 0=no arthritis and 100=extremely active arthritis), and at least 1 of 2 joint criteria with no deterioration in other criteria.
Time Frame: Weeks 16 and 24
Population: FAS1 with >=3% BSA psoriatic involvement and IGA score >=2 at baseline. Participants with both PASI 75 and modified PsARC responses at specific timepoint and did not meet TF criteria before, considered responders at that time point. Participants who met 1/more TF criteria before or with missing data at that time point considered non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 78 | 82 | 89
percentage of participants
  Week 16 | 9.0 | 48.8 | 55.1
  Week 24 | 5.1 | 50.0 | 62.9

48. Secondary Outcome: Percentage of Participants With an IGA Score of 0 (Cleared) at Weeks 16 and 24 Among the Participants With >=3% BSA Psoriatic Involvement and an IGA Score of >=2 (Mild) at Baseline
Description: The IGA documents the investigator's assessment of the patient's psoriasis and lesions are graded for induration, erythema and scaling, each using a 5 point scale: 0 (no evidence), 1 (minimal), 2 (mild), 3 (moderate), and 4 (severe). The IGA score of psoriasis was based upon the average of induration, erythema and scaling scores. The participant's psoriasis was assessed as cleared (0), minimal (1), mild (2), moderate (3), or severe (4). Participants who achieved IGA Score of 0 (cleared) at a specific timepoint and did not meet any TF criteria before, were considered as responders at that time point. Participants who met 1 or more TF criteria before or with missing data at that time point were considered as non-responders.
Time Frame: Weeks 16 and 24
Population: Analysis population is FAS1 among participants with >=3% BSA psoriatic involvement and an IGA score of >=2 at baseline.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 78 | 82 | 89
percentage of participants
  Week 16 | 9.0 | 32.9 | 40.4
  Week 24 | 7.7 | 37.8 | 53.9

49. Secondary Outcome: Change From Baseline in PASI Score at Weeks 16 and 24 Among the Participants With >=3% BSA Psoriatic Involvement and an IGA Score of >=2 (Mild) at Baseline
Description: PASI is a tool to assess and grade severity of psoriasis and response to therapy. In PASI, body is divided into 4 areas: head, trunk, upper extremities, lower extremities. Each area was assessed separately for percentage of area involved and translated to numeric score ranging from 0 (no involvement) to 6 (90 to 100% involvement), and for erythema, induration, and scaling, each rated on scale of 0 to 4 that is none to maximum severtiy. PASI numeric score range from 0 (no psoriasis) to 72. Higher scores indicate more severe disease. Negative change from baseline indicates improvement of psoriasis.
Time Frame: Baseline, Weeks 16 and 24
Population: Analysis population is FAS1 among participants who had >=3% BSA of psoriatic involvement and IGA score >=2 (mild) at baseline. Data after meeting one/more TF criteria were imputed as no change from baseline. Missing data were assumed to be MAR. LS mean is based on MMRM model that included data from all visits for all participants included in model.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 78 | 82 | 89
units on a scale
  Week 16 | -2.910 [-4.207 to -1.612] | -9.631 [-10.881 to -8.381] | -10.096 [-11.318 to -8.874]
  Week 24 | -2.317 [-3.709 to -0.926] | -9.974 [-11.323 to -8.624] | -10.915 [-12.224 to -9.605]

50. Secondary Outcome: Change From Baseline in 36-Item Short Form Health Survey (SF-36) Physical Component Summary (PCS) at Weeks 8, 16 and 24
Description: as for outcome 9
Time Frame: Baseline, Weeks 8, 16 and 24
Population: as for outcome 6
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 126 | 127 | 128
units on a scale
  Week 8 | 2.15 [1.06 to 3.23] | 2.87 [1.80 to 3.95] | 4.46 [3.39 to 5.54]
  Week 16 | 2.50 [1.31 to 3.69] | 5.26 [4.08 to 6.43] | 6.72 [5.54 to 7.89]
  Week 24 | 1.96 [0.69 to 3.24] | 6.10 [4.83 to 7.37] | 6.87 [5.60 to 8.14]

51. Secondary Outcome: Change From Baseline in 36-Item Short Form Health Survey (SF-36) Mental Component Summary (MCS) at Weeks 8, 16 and 24
Description: as for outcome 12
Time Frame: Baseline, Weeks 8, 16 and 24
Population: as for outcome 6
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 126 | 127 | 128
units on a scale
  Week 8 | 1.99 [0.73 to 3.24] | 2.72 [1.47 to 3.97] | 2.46 [1.22 to 3.71]
  Week 16 | 2.25 [0.87 to 3.63] | 2.61 [1.25 to 3.98] | 3.04 [1.68 to 4.41]
  Week 24 | 2.37 [0.93 to 3.81] | 3.20 [1.78 to 4.63] | 3.60 [2.17 to 5.02]

52. Secondary Outcome: Change From Baseline in Norm Based Scores of SF-36 Scales at Weeks 8, 16 and 24
Description: SF-36 is a multi-domain instrument with 36 items to evaluate the health status and quality of life. It included 8 subscales: physical functioning, physical role functioning, bodily pain, general health perception, vitality, social functioning, emotional role functioning, and mental health. The scores 0-100 (where higher scores indicated a better quality of life) from each subscale of SF-36 were normalized to a mean of 50 and standard deviations of 10, based upon general US population norms. Higher score indicates better health status. A positive change indicates improvement while a negative change indicates worsening of health status and quality of life.
Time Frame: Baseline, Week 8, 16 and 24
Population: as for outcome 35
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 126 | 127 | 128
units on a scale
  Week 8: Physical Function Score | 1.362 [0.201 to 2.524] | 2.616 [1.456 to 3.777] | 4.082 [2.927 to 5.237]
  Week 16: Physical Function Score | 1.901 [0.603 to 3.199] | 5.143 [3.851 to 6.434] | 6.190 [4.902 to 7.478]
  Week 24: Physical Function Score | 1.636 [0.249 to 3.023] | 5.776 [4.394 to 7.158] | 6.952 [5.571 to 8.333]
  Week 8: Role-physical Score | 2.212 [1.104 to 3.321] | 2.084 [0.978 to 3.190] | 3.834 [2.730 to 4.938]
  Week 16: Role-physical Score | 2.242 [1.037 to 3.447] | 4.224 [3.027 to 5.422] | 5.447 [4.250 to 6.644]
  Week 24: Role-physical Score | 2.319 [1.063 to 3.576] | 4.878 [3.627 to 6.130] | 5.442 [4.189 to 6.694]
  Week 8: Bodily Pain Score | 3.081 [1.876 to 4.286] | 3.886 [2.682 to 5.089] | 5.140 [3.941 to 6.338]
  Week 16: Bodily Pain Score | 3.125 [1.859 to 4.391] | 5.059 [3.800 to 6.318] | 6.778 [5.521 to 8.035]
  Week 24: Bodily Pain Score | 2.854 [1.468 to 4.240] | 6.840 [5.459 to 8.221] | 7.490 [6.110 to 8.871]
  Week 8: General Health Score | 1.989 [0.806 to 3.172] | 3.071 [1.890 to 4.252] | 3.486 [2.309 to 4.663]
  Week 16: General Health Score | 1.683 [0.492 to 2.874] | 3.769 [2.585 to 4.953] | 5.225 [4.042 to 6.408]
  Week 24: General Health Score | 1.690 [0.510 to 2.869] | 4.349 [3.175 to 5.524] | 5.174 [3.998 to 6.349]
  Week 8: Vitality Score | 2.312 [1.081 to 3.542] | 3.917 [2.689 to 5.144] | 4.614 [3.389 to 5.838]
  Week 16: Vitality Score | 3.084 [1.720 to 4.449] | 4.777 [3.422 to 6.133] | 5.589 [4.234 to 6.943]
  Week 24: Vitality Score | 2.311 [0.881 to 3.742] | 5.596 [4.172 to 7.020] | 6.426 [5.000 to 7.852]
  Week 8: Social Function Score | 2.025 [0.643 to 3.407] | 3.287 [1.907 to 4.667] | 3.798 [2.423 to 5.173]
  Week 16: Social Function Score | 2.455 [1.020 to 3.890] | 3.531 [2.105 to 4.957] | 4.817 [3.392 to 6.241]
  Week 24: Social Function Score | 2.582 [1.240 to 3.924] | 5.426 [4.089 to 6.762] | 5.227 [3.889 to 6.564]
  Week 8: Role-emotional Score | 1.980 [0.615 to 3.345] | 2.237 [0.877 to 3.598] | 1.987 [0.631 to 3.343]
  Week 16: Role-emotional Score | 1.784 [0.316 to 3.253] | 2.496 [1.040 to 3.953] | 3.265 [1.810 to 4.720]
  Week 24: Role-emotional Score | 2.201 [0.753 to 3.649] | 2.415 [0.976 to 3.853] | 3.531 [2.090 to 4.972]
  Week 8: Mental Health Score | 2.124 [0.901 to 3.348] | 2.574 [1.358 to 3.790] | 3.126 [1.914 to 4.339]
  Week 16: Mental Health Score | 2.360 [1.058 to 3.662] | 3.489 [2.200 to 4.777] | 3.984 [2.696 to 5.272]
  Week 24: Mental Health Score | 2.062 [0.658 to 3.466] | 3.818 [2.425 to 5.211] | 4.356 [2.961 to 5.751]

53. Secondary Outcome: Percentage of Participants Who Achieved >=5-point Improvement From Baseline in SF-36 MCS Score by Visit Over Time Through Week 24
Description: SF-36 is a multi-domain instrument with 36 items to evaluate the health status and quality of life. It included 8 subscales (physical functioning, physical role functioning, bodily pain, general health perception, vitality, social functioning, emotional role functioning, and mental health), which yielded a Physical Component Summary (PCS) with score range 0-100 (higher score-better quality of life) and a Mental Component Summary (MCS) with score range 0-100 (higher score-better quality of life) in addition to subscale scores. The MCS scores are normalized to a mean of 50 and standard deviations of 10, based upon general US population norms. Higher score indicates better outcome, with an increase of 5 points considered to be clinically meaningful.
Time Frame: Weeks 8, 16 and 24
Population: Analysis population is FAS1. Participants who achieved >=5-point improvement from baseline in SF-36 MCS score at specific time point and did not meet any TF criteria before, were considered as responders at that time point. Participants who met 1 or more TF criteria before or with missing data at that time point were considered as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 126 | 127 | 128
percentage of participants
  Week 8 | 27.0 | 33.9 | 35.2
  Week 16 | 31.0 | 32.3 | 39.8
  Week 24 | 25.4 | 37.8 | 43.0

54. Secondary Outcome: Percentage of Participants Who Achieved >=5 Point Improvement From Baseline in SF-36 PCS Score Through Week 24
Description: SF-36 is a multi-domain instrument with 36 items to evaluate the health status and quality of life. It included 8 subscales (physical functioning, physical role functioning, bodily pain, general health perception, vitality, social functioning, emotional role functioning, and mental health), which yielded a Physical Component Summary (PCS) with score range 0-100 (higher score-better quality of life) and a Mental Component Summary (MCS) with score range 0-100 (higher score-better quality of life) in addition to subscale scores. The PCS scores are normalized to a mean of 50 and standard deviations of 10, based upon general US population norms. Higher score indicates better outcome, with an increase of 5 points considered to be clinically meaningful.
Time Frame: Weeks 8, 16 and 24
Population: Analysis population is FAS1. Participants who achieved >=5-point improvement from baseline in SF-36 PCS score at specific time point and did not meet any TF criteria before, were considered as responders at that time point. Participants who met 1 or more TF criteria before or with missing data at that time point were considered as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 126 | 127 | 128
percentage of participants
  Week 8 | 31.0 | 33.9 | 46.1
  Week 16 | 29.4 | 48.0 | 50.0
  Week 24 | 28.6 | 51.2 | 53.9

55. Secondary Outcome: Change From Baseline in Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue Score at Weeks 8, 16, and 24
Description: The FACIT-Fatigue is a questionnaire that assesses self-reported tiredness, weakness, and difficulty conducting usual activities due to fatigue. The subscale consists 13-item instrument to measure fatigue. Each of the 13 items has a set of five response categories: Not at all (=0), A little bit (=1), Somewhat (=2), Quite a bit (=3) and Very much (=4). A total FACIT-Fatigue subscale score was calculated as the sum of the 13 item scores (reserved scores [4 - score]) and ranges from 0 to 52, with a higher score indicating less fatigue. Positive changes from baseline indicate improvement of fatigue. Items were reverse scored when appropriate to provide a scale in which higher scores represent better functioning or less fatigue.
Time Frame: Baseline, Weeks 8, 16 and 24
Population: as for outcome 35
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 126 | 127 | 128
units on a scale
  Week 8 | 2.356 [1.081 to 3.632] | 3.643 [2.369 to 4.917] | 3.576 [2.306 to 4.845]
  Week 16 | 2.164 [0.782 to 3.547] | 4.853 [3.478 to 6.228] | 4.544 [3.171 to 5.918]
  Week 24 | 2.206 [0.773 to 3.638] | 5.609 [4.181 to 7.036] | 5.841 [4.416 to 7.267]

56. Secondary Outcome: Percentage of Participants Who Achieved >=4-point Improvement From Baseline in FACIT-Fatigue Score at Weeks 8, 16, and 24
Description: The FACIT-Fatigue is a questionnaire that assesses self-reported tiredness, weakness, and difficulty conducting usual activities due to fatigue. The subscale consists 13-item instrument to measure fatigue. Each of the 13 items has a set of five response categories: Not at all (=0), A little bit (=1), Somewhat (=2), Quite a bit (=3) and Very much (=4). A total FACIT-Fatigue subscale score was calculated as the sum of the 13 item scores (reserved scores [4 - score]) and ranges from 0 to 52, with a higher score indicating less fatigue. Items were reverse scored when appropriate to provide a scale in which higher scores represent better functioning or less fatigue.
Time Frame: Weeks 8, 16, and 24
Population: Analysis population is FAS1. Participants who achieved >=4-point improvement from baseline in FACIT-fatigue score at specific time point and did not meet any TF criteria before, were considered responders at that time point. Participants who met 1 or more TF criteria before or with missing data at that time point were considered non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 126 | 127 | 128
percentage of participants
  Week 8: number analyzed (Participants) | 126 | 127 | 125
  Week 8 | 35.7 | 44.1 | 43.8
  Week 16: number analyzed (Participants) | 107 | 119 | 121
  Week 16 | 34.1 | 50.4 | 52.3
  Week 24: number analyzed (Participants) | 104 | 114 | 124
  Week 24 | 34.9 | 53.5 | 63.3

57. Secondary Outcome: Change From Baseline in Patient-Reported Outcomes Measurement Information System (PROMIS)-29 Scores at Weeks 8, 16 and 24
Description: PROMIS-29 contains 4 items for each of seven PROMIS domains (Anxiety, Depression, Fatigue, Pain Interference, Physical Function, Sleep Disturbance, and Satisfaction-Social Role and Activity. PROMIS-29 also includes an additional pain intensity 0-10 numeric rating scale (NRS). The raw score of each domain is converted into a standardized score with a mean of 50 and a standard deviation (SD) of 10 for the general population in the US (T-Score).
Time Frame: Baseline, Weeks 8, 16 and 24
Population: as for outcome 35
Measure: Least Squares Mean (95% Confidence Interval); unit: T-score
Arm/Group | Placebo | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 126 | 127 | 128
T-score
  Week 8: Anxiety | -1.98 [-3.29 to -0.66] | -2.19 [-3.50 to -0.88] | -1.83 [-3.14 to -0.53]
  Week 16: Anxiety | -2.30 [-3.63 to -0.97] | -3.08 [-4.40 to -1.75] | -2.23 [-3.54 to -0.91]
  Week 24: Anxiety | -1.37 [-2.71 to -0.03] | -3.23 [-4.57 to -1.89] | -2.92 [-4.25 to -1.59]
  Week 8: Depression | -0.86 [-2.07 to 0.35] | -2.42 [-3.63 to -1.21] | -1.54 [-2.74 to -0.34]
  Week 16: Depression | -0.85 [-2.02 to 0.31] | -2.70 [-3.87 to -1.54] | -2.69 [-3.85 to -1.54]
  Week 24: Depression | -0.85 [-2.12 to 0.42] | -3.40 [-4.66 to -2.14] | -2.67 [-3.92 to -1.41]
  Week 8: Fatigue | -1.87 [-3.13 to -0.62] | -3.25 [-4.50 to -1.99] | -2.90 [-4.14 to -1.65]
  Week 16: Fatigue | -2.29 [-3.57 to -1.02] | -4.26 [-5.53 to -2.99] | -4.14 [-5.40 to -2.88]
  Week 24: Fatigue | -1.86 [-3.24 to -0.48] | -4.79 [-6.16 to -3.42] | -5.08 [-6.45 to -3.71]
  Week 8: Pain Interference | -2.42 [-3.40 to -1.43] | -2.99 [-3.97 to -2.00] | -3.32 [-4.30 to -2.33]
  Week 16: Pain Interference | -2.62 [-3.69 to -1.55] | -3.99 [-5.06 to -2.93] | -5.02 [-6.08 to -3.96]
  Week 24: Pain Interference | -2.30 [-3.46 to -1.13] | -5.49 [-6.65 to -4.34] | -5.69 [-6.85 to -4.53]
  Week 8: Physical Function | 1.34 [0.44 to 2.23] | 1.31 [0.42 to 2.20] | 2.37 [1.48 to 3.26]
  Week 16: Physical Function | 1.53 [0.49 to 2.57] | 3.21 [2.17 to 4.24] | 4.12 [3.09 to 5.15]
  Week 24: Physical Function | 1.34 [0.25 to 2.43] | 3.89 [2.81 to 4.98] | 5.05 [3.96 to 6.13]
  Week 8: Sleep Disturbance | -1.22 [-2.23 to -0.21] | -1.91 [-2.92 to -0.91] | -2.09 [-3.09 to -1.09]
  Week 16: Sleep Disturbance | -1.54 [-2.53 to -0.54] | -3.82 [-4.82 to -2.83] | -3.09 [-4.08 to -2.10]
  Week 24: Sleep Disturbance | -1.17 [-2.25 to -0.09] | -3.48 [-4.56 to -2.40] | -2.46 [-3.53 to -1.38]
  Week 8: Satisfaction-Social Role and Activity | 1.52 [0.39 to 2.64] | 3.13 [2.01 to 4.25] | 3.18 [2.06 to 4.29]
  Week 16: Satisfaction-Social Role and Activity | 1.86 [0.65 to 3.08] | 3.93 [2.72 to 5.14] | 3.97 [2.76 to 5.17]
  Week 24: Satisfaction-Social Role and Activity | 1.45 [0.22 to 2.69] | 4.90 [3.66 to 6.13] | 4.52 [3.29 to 5.75]
  Week 8: Pain Intensity | -0.74 [-1.06 to -0.41] | -1.34 [-1.66 to -1.01] | -1.28 [-1.61 to -0.96]
  Week 16: Pain Intensity | -0.73 [-1.09 to -0.37] | -1.63 [-1.98 to -1.27] | -2.03 [-2.38 to -1.67]
  Week 24: Pain Intensity | -0.56 [-0.94 to -0.19] | -1.98 [-2.36 to -1.61] | -2.32 [-2.69 to -1.94]

58. Secondary Outcome: Change From Baseline in FACIT-Fatigue Score at Week 24 by ACR 20 Response at Week 24
Description: as for outcome 55
Time Frame: Baseline and Week 24
Population: Analysis population is FAS1. Data after meeting one or more TF criteria were imputed as no change from baseline. Here, n (number analyzed) signifies the number of participants who were ACR 20 responders or non-responders at Week 24.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 126 | 127 | 128
units on a scale
  Among ACR 20 responders: number analyzed (Participants) | 28 | 66 | 76
  Among ACR 20 responders | 8.571 (7.8995) | 9.242 (10.8473) | 6.684 (8.0948)
  Among ACR 20 non-responders: number analyzed (Participants) | 98 | 61 | 52
  Among ACR 20 non-responders | 0.316 (6.8181) | 1.984 (7.8877) | 3.635 (6.8170)

59. Secondary Outcome: Percentage of Participants Who Achieved >=4-point Improvement From Baseline in FACIT-Fatigue Score at Week 24 by ACR 20 Response at Week 24
Description: as for outcome 56
Time Frame: Week 24
Population: FAS1. Participants who achieved >=4-point improvement from baseline at Week 24 and did not meet any TF criteria before Week 24: responders. Participants who met 1 or more TF criteria or with missing data: non-responders. Here, n (number analyzed) signifies the number of participants who were ACR 20 responders or non-responders at Week 24.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 126 | 127 | 128
percentage of participants
  Among ACR 20 responders: number analyzed (Participants) | 28 | 66 | 76
  Among ACR 20 responders | 67.9 | 68.2 | 73.7
  Among ACR 20 non-responders: number analyzed (Participants) | 98 | 61 | 52
  Among ACR 20 non-responders | 25.5 | 37.7 | 48.1

60. Secondary Outcome: Percentage of Participants Who Achieved an Improvement of >=3 Points From Baseline in PROMIS-29 Domain Scores at Weeks 8, 16, and 24
Description: PROMIS-29 contains 4 items for each of seven PROMIS domains (Anxiety, Depression, Fatigue, Pain Interference, Physical Function, Sleep Disturbance, and Satisfaction-Social Role and Activity. PROMIS-29 also includes an additional pain intensity 0-10 NRS. The raw score of each domain is converted into a standardized score with a mean of 50 and a SD of 10 for the general population in the US (T-Score).
Time Frame: Weeks 8, 16, and 24
Population: Analysis population is FAS1. Participants who achieved >=3-point improvement from baseline in PROMIS-29 domain scores at a specific timepoint and did not meet any TF criteria before, considered as responders at that time point. Participants who met 1 or more TF criteria before or with missing data at that time point, considered as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 126 | 127 | 128
percentage of participants
  Week 8: Anxiety | 41.3 | 41.7 | 39.1
  Week 16: Anxiety | -34.9 | 42.5 | 41.4
  Week 24: Anxiety | 34.9 | 45.7 | 42.2
  Week 8: Depression | 24.6 | 30.7 | 34.4
  Week 16: Depression | 25.4 | 35.4 | 33.6
  Week 24: Depression | 26.2 | 39.4 | 38.3
  Week 8: Fatigue | 34.1 | 39.4 | 42.2
  Week 16: Fatigue | 38.9 | 49.6 | 49.2
  Week 24: Fatigue | 32.5 | 48.8 | 55.5
  Week 8: Pain Interference | 34.9 | 41.7 | 43.8
  Week 16: Pain Interference | 39.7 | 47.2 | 56.3
  Week 24: Pain Interference | 33.3 | 54.3 | 57.0
  Week 8: Physical Function | 28.6 | 30.7 | 40.6
  Week 16: Physical Function | 28.6 | 44.1 | 45.3
  Week 24: Physical Function | 22.2 | 48.0 | 53.9
  Week 8: Sleep Disturbance | 35.7 | 38.6 | 39.1
  Week 16: Sleep Disturbance | 36.5 | 48.8 | 38.3
  Week 24: Sleep Disturbance | 31.0 | 48.8 | 40.6
  Week 8: Satisfaction-Social Role and Activity | 35.7 | 44.9 | 49.2
  Week 16: Satisfaction-Social Role and Activity | 37.3 | 46.5 | 46.1
  Week 24: Satisfaction-Social Role and Activity | 32.5 | 52.0 | 50.0
  Week 8: Pain Intensity | 15.1 | 22.8 | 26.6
  Week 16: Pain Intensity | 18.3 | 33.1 | 42.2
  Week 24: Pain Intensity | 15.1 | 37.0 | 45.3

61. Secondary Outcome: Percentage of Participants Who Achieved an Improvement of >=5 Points From Baseline in PROMIS-29 Domain Scores at Weeks 8, 16, and 24
Description: as for outcome 60
Time Frame: Weeks 8, 16, and 24
Population: Analysis population is FAS1. Participants who achieved >=5-point improvement from baseline in PROMIS-29 domain scores at a specific timepoint and did not meet any TF criteria before, considered as responders at that time point. Participants who met 1 or more TF criteria before or with missing data at that time point, considered as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 126 | 127 | 128
percentage of participants
  Week 8: Anxiety | 33.3 | 37.0 | 29.7
  Week 16: Anxiety | 29.4 | 34.6 | 33.6
  Week 24: Anxiety | 28.6 | 41.7 | 38.3
  Week 8: Depression | 17.5 | 27.6 | 26.6
  Week 16: Depression | 19.0 | 32.3 | 28.9
  Week 24: Depression | 19.8 | 36.2 | 30.5
  Week 8: Fatigue | 27.8 | 29.1 | 33.6
  Week 16: Fatigue | 33.3 | 40.9 | 43.0
  Week 24: Fatigue | 31.0 | 45.7 | 47.7
  Week 8: Pain Interference | 22.2 | 29.9 | 35.9
  Week 16: Pain Interference | 29.4 | 38.6 | 43.8
  Week 24: Pain Interference | 23.8 | 46.5 | 51.6
  Week 8: Physical Function | 15.1 | 18.9 | 22.7
  Week 16: Physical Function | 18.3 | 26.8 | 32.8
  Week 24: Physical Function | 15.9 | 36.2 | 39.8
  Week 8: Sleep Disturbance | 24.6 | 24.4 | 27.3
  Week 16: Sleep Disturbance | 24.6 | 40.2 | 30.5
  Week 24: Sleep Disturbance | 21.4 | 37.0 | 32.8
  Week 8: Satisfaction-Social Role and Activity | 25.4 | 40.2 | 38.3
  Week 16: Satisfaction-Social Role and Activity | 30.2 | 42.5 | 39.8
  Week 24: Satisfaction-Social Role and Activity | 22.2 | 45.7 | 43.0
  Week 8: Pain Intensity | 5.6 | 6.3 | 6.3
  Week 16: Pain Intensity | 6.3 | 8.7 | 14.8
  Week 24: Pain Intensity | 4.0 | 18.1 | 18.0

62. Secondary Outcome: Percentage of Participants Who Achieved ACR 20 Response at Weeks 24, 28, 36, 44 and 52
Description: as for outcome 15
Time Frame: Weeks 24, 28, 36, 44 and 52
Population: Analysis population is full analysis set 2 (FAS2) included all randomized participants who were still on study treatment at Week 24. Here, n (number analyzed) signifies the number of participants analyzed at specified timepoints.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 114 | 123 | 125
percentage of participants
  Week 24 | 27.2 | 54.5 | 60.8
  Week 28: number analyzed (Participants) | 112 | 122 | 125
  Week 28 | 50.0 | 68.9 | 74.4
  Week 36: number analyzed (Participants) | 109 | 118 | 121
  Week 36 | 56.9 | 70.3 | 71.1
  Week 44: number analyzed (Participants) | 107 | 117 | 125
  Week 44 | 61.7 | 73.5 | 72.0
  Week 52: number analyzed (Participants) | 104 | 112 | 124
  Week 52 | 68.3 | 67.9 | 75.8

63. Secondary Outcome: Percentage of Participants Who Achieved ACR 50 Response at Weeks 24, 28, 36, 44 and 52
Description: as for outcome 16
Time Frame: Weeks 24, 28, 36, 44 and 52
Population: Analysis population is FAS2. Here, n (number analyzed) signifies the number of participants analyzed at specified timepoints.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 114 | 123 | 125
percentage of participants
  Week 24 | 9.6 | 30.9 | 36.8
  Week 28: number analyzed (Participants) | 112 | 122 | 125
  Week 28 | 21.4 | 42.6 | 39.2
  Week 36: number analyzed (Participants) | 110 | 119 | 121
  Week 36 | 32.7 | 47.1 | 44.6
  Week 44: number analyzed (Participants) | 107 | 117 | 124
  Week 44 | 30.8 | 51.3 | 46.0
  Week 52: number analyzed (Participants) | 104 | 113 | 124
  Week 52 | 36.5 | 43.4 | 55.6

64. Secondary Outcome: Percentage of Participants Who Achieved ACR 70 Response at Weeks 24, 28, 36, 44 and 52
Description: ACR 70 response was defined as >=70% improvement from baseline in both swollen joint count (66 joints) and tender joint count (68 joints), and >=70% improvement from baseline in 3 of the 5 assessments: patient's assessment of pain using VAS (0-100 mm, 0=no pain and 100=worst possible pain), patient's global assessment of disease activity (arthritis, VAS; 0-100 mm, 0=excellent and 100= poor), physician's global assessment of disease activity (VAS; 0-100 mm, 0=no arthritis activity and 100=extremely active arthritis), patient's assessment of physical function measured by HAQ-DI (defined as a 20-question instrument assessing 8 functional areas; range: 0-3, 0=indicating no difficulty, 3=indicating inability to perform a task in that area), and CRP.
Time Frame: Weeks 24, 28, 36, 44 and 52
Population: as for outcome 63
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 114 | 123 | 125
percentage of participants
  Week 24 | 6.1 | 12.2 | 20.8
  Week 28: number analyzed (Participants) | 112 | 122 | 125
  Week 28 | 9.8 | 20.5 | 24.8
  Week 36: number analyzed (Participants) | 111 | 119 | 121
  Week 36 | 18.0 | 25.2 | 26.4
  Week 44: number analyzed (Participants) | 107 | 116 | 125
  Week 44 | 16.8 | 28.4 | 26.4
  Week 52: number analyzed (Participants) | 104 | 114 | 124
  Week 52 | 19.2 | 28.9 | 29.8

65. Secondary Outcome: Percent Change From Baseline in ACR Components at Weeks 24, 28, 36, 44 and 52
Description: as for outcome 22
Time Frame: Baseline, Weeks 24, 28, 36, 44 and 52
Population: as for outcome 63
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 114 | 123 | 125
percent change
  Week 24: Swollen Joint Count | -48.33 (45.987) | -66.62 (47.086) | -73.23 (38.120)
  Week 28: Swollen Joint Count: number analyzed (Participants) | 112 | 123 | 125
  Week 28: Swollen Joint Count | -59.95 (47.826) | -75.42 (33.774) | -80.93 (27.197)
  Week 36: Swollen Joint Count: number analyzed (Participants) | 111 | 119 | 122
  Week 36: Swollen Joint Count | -70.50 (37.359) | -79.16 (35.141) | -80.19 (29.160)
  Week 44: Swollen Joint Count: number analyzed (Participants) | 108 | 117 | 125
  Week 44: Swollen Joint Count | -72.63 (38.625) | -80.35 (34.653) | -82.46 (31.652)
  Week 52: Swollen Joint Count: number analyzed (Participants) | 103 | 112 | 124
  Week 52: Swollen Joint Count | -78.23 (37.345) | -79.63 (36.471) | -86.73 (26.776)
  Week 24: Tender Joint Count | -27.58 (53.737) | -53.73 (45.118) | -56.56 (41.774)
  Week 28: Tender Joint Count: number analyzed (Participants) | 112 | 123 | 125
  Week 28: Tender Joint Count | -42.99 (62.128) | -64.03 (40.678) | -66.68 (31.528)
  Week 36: Tender Joint Count: number analyzed (Participants) | 111 | 119 | 122
  Week 36: Tender Joint Count | -57.06 (43.351) | -68.44 (39.771) | -64.67 (41.606)
  Week 44: Tender Joint Count: number analyzed (Participants) | 108 | 117 | 125
  Week 44: Tender Joint Count | -60.08 (42.811) | -69.23 (51.229) | -71.90 (31.422)
  Week 52: Tender Joint Count: number analyzed (Participants) | 103 | 112 | 124
  Week 52: Tender Joint Count | -65.65 (37.682) | -72.39 (35.102) | -72.70 (37.487)
  Week 24: Patient's Assessment of Pain: number analyzed (Participants) | 113 | 123 | 124
  Week 24: Patient's Assessment of Pain | -6.05 (52.682) | -32.65 (45.343) | -38.90 (43.955)
  Week 28: Patient's Assessment of Pain: number analyzed (Participants) | 110 | 122 | 124
  Week 28: Patient's Assessment of Pain | -21.93 (52.597) | -38.86 (45.149) | -43.59 (39.524)
  Week 36: Patient's Assessment of Pain: number analyzed (Participants) | 109 | 120 | 120
  Week 36: Patient's Assessment of Pain | -27.61 (56.373) | -42.85 (43.952) | -47.23 (41.167)
  Week 44: Patient's Assessment of Pain: number analyzed (Participants) | 107 | 117 | 124
  Week 44: Patient's Assessment of Pain | -27.98 (64.080) | -45.27 (47.794) | -48.97 (36.509)
  Week 52: Patient's Assessment of Pain: number analyzed (Participants) | 103 | 114 | 123
  Week 52: Patient's Assessment of Pain | -35.64 (66.672) | -42.67 (47.250) | -50.03 (50.203)
  Week 24: PtGA of Disease Activity | -7.63 (58.147) | -37.16 (39.760) | -40.27 (42.250)
  Week 28: PtGA of Disease Activity: number analyzed (Participants) | 111 | 122 | 125
  Week 28: PtGA of Disease Activity | -21.74 (57.662) | -45.35 (41.564) | -37.62 (60.121)
  Week 36: PtGA of Disease Activity: number analyzed (Participants) | 110 | 120 | 121
  Week 36: PtGA of Disease Activity | -26.51 (60.926) | -46.03 (39.547) | -45.17 (39.277)
  Week 44: PtGA of Disease Activity: number analyzed (Participants) | 108 | 117 | 125
  Week 44: PtGA of Disease Activity | -21.76 (81.481) | -46.11 (40.973) | -45.84 (43.368)
  Week 52: PtGA of Disease Activity: number analyzed (Participants) | 103 | 114 | 124
  Week 52: PtGA of Disease Activity | -35.17 (56.398) | -45.84 (42.176) | -47.85 (55.429)
  Week 24: PGA of Disease Activity: number analyzed (Participants) | 113 | 122 | 125
  Week 24: PGA of Disease Activity | -33.22 (34.014) | -53.43 (37.305) | -61.59 (31.445)
  Week 28: PGA of Disease Activity: number analyzed (Participants) | 111 | 122 | 123
  Week 28: PGA of Disease Activity | -53.88 (31.619) | -57.70 (33.724) | -65.96 (29.400)
  Week 36: PGA of Disease Activity: number analyzed (Participants) | 109 | 117 | 120
  Week 36: PGA of Disease Activity | -62.40 (29.215) | -64.51 (34.389) | -68.37 (27.206)
  Week 44: PGA of Disease Activity: number analyzed (Participants) | 107 | 117 | 124
  Week 44: PGA of Disease Activity | -64.93 (28.895) | -69.08 (30.743) | -72.65 (25.842)
  Week 52: PGA of Disease Activity: number analyzed (Participants) | 103 | 111 | 124
  Week 52: PGA of Disease Activity | -68.67 (32.861) | -68.83 (32.776) | -74.71 (25.456)
  Week 24: HAQ-DI score: number analyzed (Participants) | 108 | 121 | 118
  Week 24: HAQ-DI score | -7.65 (62.206) | -8.80 (148.199) | -31.18 (72.701)
  Week 28: HAQ-DI score: number analyzed (Participants) | 105 | 121 | 118
  Week 28: HAQ-DI score | -15.62 (51.720) | -29.10 (60.044) | -33.41 (72.942)
  Week 36: HAQ-DI score: number analyzed (Participants) | 104 | 118 | 114
  Week 36: HAQ-DI score | -15.37 (53.391) | -29.43 (73.712) | -32.74 (86.404)
  Week 44: HAQ-DI score: number analyzed (Participants) | 102 | 116 | 118
  Week 44: HAQ-DI score | -29.61 (45.603) | -34.54 (73.685) | -35.91 (80.885)
  Week 52: HAQ-DI score: number analyzed (Participants) | 100 | 112 | 117
  Week 52: HAQ-DI score | -28.42 (45.473) | -31.09 (60.232) | -46.13 (56.354)
  Week 24: CRP: number analyzed (Participants) | 114 | 122 | 125
  Week 24: CRP | -13.58 (150.494) | -7.83 (101.789) | -6.48 (149.288)
  Week 28: CRP: number analyzed (Participants) | 111 | 121 | 124
  Week 28: CRP | -8.67 (122.851) | -5.58 (99.590) | -10.30 (97.703)
  Week 36: CRP: number analyzed (Participants) | 112 | 119 | 124
  Week 36: CRP | -17.33 (102.168) | -31.55 (50.560) | -14.65 (113.746)
  Week 44: CRP: number analyzed (Participants) | 107 | 116 | 124
  Week 44: CRP | -29.10 (70.460) | -17.81 (76.247) | -4.39 (190.368)
  Week 52: CRP: number analyzed (Participants) | 106 | 117 | 123
  Week 52: CRP | -1.68 (167.086) | -19.28 (69.875) | -15.76 (129.101)

66. Secondary Outcome: Change From Baseline in HAQ-DI Score at Weeks 24, 28, 36, 44 and 52
Description: as for outcome 2
Time Frame: Baseline, Weeks 24, 28, 36, 44 and 52
Population: as for outcome 63
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 114 | 123 | 125
units on a scale
  Week 24 | -0.1217 (0.52442) | -0.3374 (0.56967) | -0.3740 (0.45914)
  Week 28: number analyzed (Participants) | 111 | 123 | 125
  Week 28 | -0.2241 (0.50876) | -0.4004 (0.52303) | -0.3850 (0.46381)
  Week 36: number analyzed (Participants) | 110 | 120 | 121
  Week 36 | -0.2602 (0.51278) | -0.4396 (0.54426) | -0.4132 (0.47155)
  Week 44: number analyzed (Participants) | 108 | 118 | 125
  Week 44 | -0.3634 (0.53486) | -0.4672 (0.57140) | -0.4180 (0.51394)
  Week 52: number analyzed (Participants) | 104 | 114 | 124
  Week 52 | -0.3642 (0.51084) | -0.4364 (0.56400) | -0.4970 (0.47990)

67. Secondary Outcome: Percentage of Participants Who Achieved a Clinically Meaningful Improvement (>=0.35 Improvement From Baseline) in HAQ-DI Score at Weeks 24, 28, 36, 44 and 52 Among Participants With HAQ-DI Score >=0.35 at Baseline
Description: HAQ-DI score assess functional status of participant. It is 20 question instrument that assess degree of difficulty a person has in accomplishing tasks in 8 functional areas (dressing, arising, eating, walking, hygiene, reaching, gripping, and activities of daily living). Responses in each functional area were scored from 0=indicating no difficulty, to 3=indicating inability to perform a task in that area. Total HAQ score is average of the computed categories scores ranging from 0-3 where 0=least difficulty and 3=extreme difficulty. Lower scores are indicative of better functioning and a decrease of 0.35 from baseline in HAQ-DI score indicates a meaningful improvement.
Time Frame: Weeks 24, 28, 36, 44 and 52
Population: Analysis population is FAS2 among participants with HAQ-DI score >=0.35 at baseline. Here, n (number analyzed) signifies the number of participants analyzed at specified timepoints.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 100 | 109 | 109
percentage of participants
  Week 24 | 36.0 | 53.2 | 57.8
  Week 28: number analyzed (Participants) | 97 | 109 | 109
  Week 28 | 40.2 | 61.5 | 61.5
  Week 36: number analyzed (Participants) | 96 | 106 | 105
  Week 36 | 41.7 | 60.4 | 61.9
  Week 44: number analyzed (Participants) | 94 | 104 | 109
  Week 44 | 50.0 | 58.7 | 62.4
  Week 52: number analyzed (Participants) | 92 | 101 | 108
  Week 52 | 54.3 | 57.4 | 68.5

68. Secondary Outcome: Change From Baseline in DAS28 (CRP) Score at Weeks 24, 28, 36, 44 and 52
Description: DAS28 based on CRP is an index combining tender joints (28 joints), swollen joints (28 joints), CRP and patient's global assessment of disease activity. The set of 28 joint count is based on evaluation of the shoulder, elbow, wrist, metacarpophalangeal (MCP) MCP1 to MCP5, proximal interphalangeal (PIP) PIP1 to PIP5 joints of both the upper right extremity and the upper left extremity as well as the knee joints of lower right and lower left extremities. The values are 0=best to 10=worst. Negative changes from baseline indicate improvement of arthritis.
Time Frame: Baseline, Weeks 24, 28, 36, 44 and 52
Population: as for outcome 63
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 114 | 123 | 125
units on a scale
  Week 24: number analyzed (Participants) | 114 | 122 | 125
  Week 24 | -0.84 (1.043) | -1.49 (1.140) | -1.57 (1.045)
  Week 28: number analyzed (Participants) | 110 | 120 | 124
  Week 28 | -1.33 (1.121) | -1.71 (1.126) | -1.67 (1.020)
  Week 36: number analyzed (Participants) | 110 | 118 | 121
  Week 36 | -1.60 (1.123) | -1.96 (1.145) | -1.78 (1.054)
  Week 44: number analyzed (Participants) | 105 | 114 | 124
  Week 44 | -1.69 (1.224) | -1.96 (1.226) | -1.92 (1.116)
  Week 52: number analyzed (Participants) | 103 | 112 | 123
  Week 52 | -1.84 (1.087) | -2.03 (1.250) | -1.99 (1.062)

69. Secondary Outcome: Percentage of Participants Who Achieved a DAS28 (CRP) Response at Weeks 24, 28, 36, 44 and 52
Description: DAS28 based on CRP is an index combining tender joints (28 joints), swollen joints (28 joints), CRP and patient's global assessment of disease activity. The set of 28 joint count is based on evaluation of the shoulder, elbow, wrist, metacarpophalangeal (MCP) MCP1 to MCP5, proximal interphalangeal (PIP) PIP1 to PIP5 joints of both the upper right extremity and the upper left extremity as well as the knee joints of lower right and lower left extremities. DAS28 (CRP) response criteria was defined as follows: Good response: <=3.2 at visit and >1.2 improvement; Moderate response: >3.2 at visit and >1.2 improvement or <=5.1 at visit and >0.6-1.2 improvement; No response: <=0.6 improvement, or >5.1 at visit and <=1.2 improvement. The values are 0=best to 10=worst. A DAS28 (CRP) responder was defined as achieving a good or moderate DAS28 response at a specific visit.
Time Frame: Weeks 24, 28, 36, 44 and 52
Population: as for outcome 63
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 114 | 123 | 125
percentage of participants
  Week 24: number analyzed (Participants) | 114 | 122 | 125
  Week 24 | 51.8 | 74.6 | 78.4
  Week 28: number analyzed (Participants) | 110 | 120 | 124
  Week 28 | 73.6 | 83.3 | 83.9
  Week 36: number analyzed (Participants) | 110 | 118 | 121
  Week 36 | 76.4 | 89.0 | 86.8
  Week 44: number analyzed (Participants) | 105 | 114 | 124
  Week 44 | 80.0 | 86.8 | 89.5
  Week 52: number analyzed (Participants) | 103 | 112 | 121
  Week 52 | 86.4 | 88.4 | 87.8

70. Secondary Outcome: Percentage of Participants Who Achieved a DAS28 (CRP) Remission at Weeks 24, 28, 36, 44 and 52
Description: DAS28 based on CRP is an index combining tender joints (28 joints), swollen joints (28 joints), CRP and patient's global assessment of disease activity. The set of 28 joint count is based on evaluation of the shoulder, elbow, wrist, metacarpophalangeal (MCP) MCP1 to MCP5, proximal interphalangeal (PIP) PIP1 to PIP5 joints of both the upper right extremity and the upper left extremity as well as the knee joints of lower right and lower left extremities. The values are 0=best to 10=worst. DAS28 (CRP) remission was defined as DAS28 (CRP) value <2.6 at the analysis visit.
Time Frame: Weeks 24, 28, 36, 44 and 52
Population: as for outcome 63
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 114 | 123 | 125
percentage of participants
  Week 24: number analyzed (Participants) | 114 | 122 | 125
  Week 24 | 14.9 | 24.6 | 36.8
  Week 28: number analyzed (Participants) | 110 | 120 | 124
  Week 28 | 26.4 | 37.5 | 38.7
  Week 36: number analyzed (Participants) | 110 | 118 | 121
  Week 36 | 39.1 | 40.7 | 40.5
  Week 44: number analyzed (Participants) | 105 | 114 | 124
  Week 44 | 38.1 | 45.6 | 51.6
  Week 52: number analyzed (Participants) | 103 | 112 | 123
  Week 52 | 37.9 | 43.8 | 56.1

71. Secondary Outcome: Percentage of Participants Who Maintained a HAQ-DI Response (>=0.35 Improvement From Baseline in HAQ-DI Score) at Week 52 Among Participants Who Achieved a HAQ-DI Response at Week 24
Description: as for outcome 67
Time Frame: Week 52
Population: Analysis population is FAS2 among participants who achieved a HAQ-DI response at Week 24. The outcome measure (OM) was planned to assess the maintenance of guselkumab effect only through Week 52, hence the data in this outcome measure is reported for guselkumab 100 mg q8w and guselkumab 100 mg q4w arms only and not for placebo arm.
Measure: Number; unit: percentage of participants
Arm/Group | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 53 | 63
percentage of participants | 84.9 | 87.3

72. Secondary Outcome: Percentage of Participants Who Achieved a Response Based on Modified Psoriatic Arthritis Responder Criteria (PsARC) at Weeks 24, 28, 36, 44 and 52
Description: The modified PsARC response was defined as improvement in at least 2 of the four criteria: >=30% decrease in swollen joint count, >=30% decrease in tender joint count, >=20% improvement in patient's Global Assessment of Disease Activity (arthritis) on a VAS (0-100 mm, 0=excellent and 100= poor), >=20% improvement in physician's Global Assessment of Disease Activity using VAS (VAS: 0-100 mm, 0=no arthritis activity and 100=extremely active arthritis), and at least one of the 2 joint criteria with no deterioration in the other criteria.
Time Frame: Weeks 24, 28, 36, 44 and 52
Population: as for outcome 63
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 114 | 123 | 125
percentage of participants
  Week 24: number analyzed (Participants) | 113 | 122 | 125
  Week 24 | 37.2 | 63.1 | 74.4
  Week 28: number analyzed (Participants) | 111 | 122 | 124
  Week 28 | 64.9 | 78.7 | 82.3
  Week 36: number analyzed (Participants) | 109 | 118 | 120
  Week 36 | 68.8 | 80.5 | 80.0
  Week 44: number analyzed (Participants) | 107 | 116 | 125
  Week 44 | 73.8 | 81.9 | 80.0
  Week 52: number analyzed (Participants) | 103 | 111 | 124
  Week 52 | 73.8 | 83.8 | 83.9

73. Secondary Outcome: Change From Baseline in the Disease Activity Index for Psoriatic Arthritis (DAPSA) Score at Weeks 24, 28, 36, 44 and 52
Description: DAPSA assessed the joint domain of PsA and was derived from the sum of the following components: tender joint count (0-68), swollen joint count (0-66), CRP level (mg/dL), patient assessment of pain (0-10cm VAS, 0=no pain, 10=worst possible pain), and patient's global assessment of disease activity on arthritis (0 to 10cm VAS, 0=excellent and 10=poor). A higher score indicates more active disease activity. Negative changes from baseline indicate improvement of PsA disease activity. The assessment does not have a score range with an upper or lower bound.
Time Frame: Baseline, Weeks 24, 28, 36, 44 and 52
Population: as for outcome 63
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 114 | 123 | 125
units on a scale
  Week 24: number analyzed (Participants) | 114 | 122 | 125
  Week 24 | -12.962 (17.9137) | -23.373 (20.2784) | -20.530 (13.2678)
  Week 28: number analyzed (Participants) | 110 | 120 | 124
  Week 28 | -18.632 (19.4997) | -26.790 (19.3655) | -22.766 (12.8366)
  Week 36: number analyzed (Participants) | 110 | 118 | 121
  Week 36 | -22.360 (18.8976) | -30.070 (21.0899) | -24.067 (14.0976)
  Week 44: number analyzed (Participants) | 105 | 114 | 124
  Week 44 | -23.602 (19.9198) | -30.312 (22.5854) | -26.010 (15.3230)
  Week 52: number analyzed (Participants) | 103 | 112 | 123
  Week 52 | -26.058 (18.6507) | -30.906 (23.0188) | -26.562 (15.1985)

74. Secondary Outcome: Percentage of Participants Who Achieved Both PASI 75 and Modified PsARC Response at Weeks 24 and 52 Among Participants With >=3% BSA Psoriatic Involvement and an IGA Score of >=2 at Baseline
Description: In PASI, each area (head, trunk, upper and lower extremities) was assessed separately for % of area involved and translated to numeric score ranging from 0 (no involvement) to 6 (90-100% involvement), and for erythema, induration, and scaling, each rated on scale of 0 to 4. PASI produces numeric score range from 0 to 72. Higher scores=more severe disease. PASI75 response: >=75% improvement in PASI score from baseline. Modified PsARC response: improvement in at least 2 of 4 criteria: >=30% decrease in SJC and TJC, >=20% improvement in PtGA of Disease Activity (arthritis) on VAS (0-100 mm, 0=excellent and 100=poor), >=20% improvement in PGA of Disease Activity on VAS (VAS: 0-100 mm, 0=no arthritis and 100=extremely active arthritis), and at least 1 of 2 joint criteria with no deterioration in other criteria.
Time Frame: Weeks 24 and 52
Population: Analysis population is FAS2 among the participants who had >=3% BSA of psoriatic involvement and an IGA score >=2 (mild) at baseline. Here, n (number analyzed) signifies the number of participants analyzed at specified timepoints.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 68 | 82 | 88
percentage of participants
  Week 24: number analyzed (Participants) | 68 | 81 | 88
  Week 24 | 8.8 | 50.6 | 63.6
  Week 52: number analyzed (Participants) | 65 | 75 | 88
  Week 52 | 69.2 | 70.7 | 79.5

75. Secondary Outcome: Percentage of Participants Who Achieved Both PASI 75 and ACR 20 Responses at Weeks 24 and 52 Among Participants With >=3% BSA Psoriatic Involvement and an IGA Score of >=2 at Baseline
Description: In PASI, each area (head, trunk, upper and lower extremities) was assessed for % of area involved and translated to numeric score from 0 (no involvement) to 6 (90-100% involvement) and for erythema, induration, and scaling, each rated on scale of 0 to 4. PASI produces numeric score from 0 to 72. Higher scores=more severe disease. PASI 75: >=75% improvement in PASI score from baseline. ACR 20: >=20% improvement in SJC (66 joints)+TJC (68 joints) and >=20% improvement in 3 of 5: patient's assessment of pain (VAS; 0-100 mm, 0=no pain to 100=worst possible pain), PtGA of disease activity (VAS; 0-100 mm, 0=excellent to 100=poor), PGA of disease activity (VAS; 0-100 mm, 0=no arthritis to 100=extremely active arthritis), patient's assessment of physical function (HAQ-DI -20-question instrument; range- 0=no difficulty to 3=inability to perform task) and CRP.
Time Frame: Weeks 24 and 52
Population: as for outcome 74
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 68 | 82 | 88
percentage of participants
  Week 24: number analyzed (Participants) | 68 | 81 | 88
  Week 24 | 10.3 | 40.7 | 53.4
  Week 52: number analyzed (Participants) | 65 | 75 | 88
  Week 52 | 64.6 | 58.7 | 73.9

76. Secondary Outcome: Change From Baseline in PASI Score at Weeks 24 and 52 Among Participants With >=3% BSA Psoriatic Involvement and an IGA Score of >=2 at Baseline
Description: PASI is a tool to assess and grade severity of psoriasis and response to therapy. In PASI, body is divided into 4 areas: head, trunk, upper extremities, lower extremities. Each area was assessed separately for percentage of area involved and translated to numeric score ranging from 0 (no involvement) to 6 (90 to 100% involvement), and for erythema, induration, and scaling, each rated on scale of 0 to 4 that is none to maximum severity. PASI numeric score range from 0 (no psoriasis) to 72. Higher scores indicate more severe disease. Negative changes from baseline indicate improvement of psoriasis.
Time Frame: Baseline, Weeks 24 and 52
Population: as for outcome 74
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 68 | 82 | 88
units on a scale
  Week 24: number analyzed (Participants) | 68 | 81 | 88
  Week 24 | -3.046 (9.3053) | -9.968 (10.0178) | -11.614 (10.3771)
  Week 52: number analyzed (Participants) | 66 | 75 | 88
  Week 52 | -10.565 (8.8792) | -10.431 (11.0277) | -11.988 (10.3067)

77. Secondary Outcome: Percentage of Participants Who Achieved PASI 75 Response at Weeks 24 and 52 Among Participants With >=3% BSA Psoriatic Involvement and an IGA Score of >=2 at Baseline
Description: PASI is a tool to assess and grade severity of psoriasis and response to therapy. In PASI, body is divided into 4 areas: head, trunk, upper extremities, lower extremities. Each area was assessed separately for percentage of area involved and translated to numeric score ranging from 0 (no involvement) to 6 (90 to 100% involvement), and for erythema, induration, and scaling, each rated on scale of 0 to 4 that is none to maximum severity. PASI numeric score range from 0 (no psoriasis) to 72. Higher scores indicate more severe disease. PASI 75 response: >=75% improvement in PASI score from baseline.
Time Frame: Weeks 24 and 52
Population: as for outcome 74
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 68 | 82 | 88
percentage of participants
  Week 24: number analyzed (Participants) | 68 | 81 | 88
  Week 24 | 20.6 | 76.5 | 87.5
  Week 52: number analyzed (Participants) | 66 | 75 | 88
  Week 52 | 84.8 | 80.0 | 94.3

78. Secondary Outcome: Percentage of Participants Who Achieved PASI 90 Response at Weeks 24 and 52 Among Participants With >=3% BSA Psoriatic Involvement and an IGA Score of >=2 at Baseline
Description: PASI is a tool to assess and grade severity of psoriasis and response to therapy. In PASI, body is divided into 4 areas: head, trunk, upper extremities, lower extremities. Each area was assessed separately for percentage of area involved and translated to numeric score ranging from 0 (no involvement) to 6 (90 to 100% involvement), and for erythema, induration, and scaling, each rated on scale of 0 to 4 that is none to maximum severity. PASI numeric score range from 0 (no psoriasis) to 72. Higher scores indicate more severe disease. PASI 90 response: >=90% improvement in PASI score from baseline.
Time Frame: Weeks 24 and 52
Population: as for outcome 74
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 68 | 82 | 88
percentage of participants
  Week 24: number analyzed (Participants) | 68 | 81 | 88
  Week 24 | 13.2 | 50.6 | 63.6
  Week 52: number analyzed (Participants) | 66 | 75 | 88
  Week 52 | 72.7 | 66.7 | 76.1

79. Secondary Outcome: Percentage of Participants Who Achieved PASI 100 Response at Weeks 24 and 52 Among Participants With >=3% BSA Psoriatic Involvement and an IGA Score of >=2 at Baseline
Description: PASI is a tool to assess and grade severity of psoriasis and response to therapy. In PASI, body is divided into 4 areas: head, trunk, upper extremities, lower extremities. Each area was assessed separately for percentage of area involved and translated to numeric score ranging from 0 (no involvement) to 6 (90 to 100% involvement), and for erythema, induration, and scaling, each rated on scale of 0 to 4 that is none to maximum severity. PASI numeric score range from 0 (no psoriasis) to 72. Higher scores indicate more severe disease. PASI 100 response: 100% improvement in PASI score from baseline.
Time Frame: Weeks 24 and 52
Population: as for outcome 74
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 68 | 82 | 88
percentage of participants
  Week 24: number analyzed (Participants) | 68 | 81 | 88
  Week 24 | 7.4 | 25.9 | 45.5
  Week 52: number analyzed (Participants) | 66 | 75 | 88
  Week 52 | 62.1 | 48.0 | 64.8

80. Secondary Outcome: Percentage of Participants Who Achieved >=5 Point Improvement From Baseline in SF-36 PCS Score at Weeks 24, 36 and 52
Description: as for outcome 54
Time Frame: Weeks 24, 36 and 52
Population: as for outcome 63
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 114 | 123 | 125
percentage of participants
  Week 24: number analyzed (Participants) | 114 | 123 | 124
  Week 24 | 35.1 | 53.7 | 55.6
  Week 36: number analyzed (Participants) | 107 | 119 | 120
  Week 36 | 44.9 | 53.8 | 55.0
  Week 52: number analyzed (Participants) | 104 | 114 | 124
  Week 52 | 52.9 | 53.5 | 62.9

81. Secondary Outcome: Percentage of Participants Who Achieved >=5 Point Improvement From Baseline in SF-36 MCS Score at Weeks 24, 36 and 52
Description: as for outcome 53
Time Frame: Weeks 24, 36 and 52
Population: as for outcome 63
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 114 | 123 | 125
percentage of participants
  Week 24: number analyzed (Participants) | 114 | 123 | 124
  Week 24 | 29.8 | 39.0 | 44.4
  Week 36: number analyzed (Participants) | 107 | 119 | 120
  Week 36 | 39.3 | 39.5 | 49.2
  Week 52: number analyzed (Participants) | 104 | 114 | 124
  Week 52 | 37.5 | 46.5 | 47.6

82. Secondary Outcome: Percentage of Participants Who Achieved Minimal Disease Activity (MDA) at Weeks 24 and 52
Description: MDA is a measure that defines a satisfactory state of disease activity that includes the 5 domains of PsA (joint symptoms, skin psoriasis, patient's perspective of pain and disease activity, physical function, and enthesitis). A participant was considered as having achieved the PsA MDA at a visit if the participant has fulfilled at least 5 of the following 7 criteria at that visit: Tender joint count (68 joints)<=1, Swollen joint count (66 joints) <=1, Psoriasis activity and severity index <=1, Patient's Assessment of Pain <=15 on a 100-unit VAS, Patient's Global Assessment of Disease Activity (arthritis and psoriasis) <=20 on a 100-unit VAS, HAQ-DI score <=0.5, and Tender entheseal points <= 1 (LEI index score <= 1).
Time Frame: Weeks 24 and 52
Population: as for outcome 63
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 114 | 123 | 125
percentage of participants
  Week 24 | 12.3 | 23.6 | 31.2
  Week 52: number analyzed (Participants) | 103 | 112 | 124
  Week 52 | 31.1 | 33.9 | 40.3

83. Secondary Outcome: Change From Baseline in Group of Research and Assessment of Psoriasis and Psoriatic Arthritis Composite (GRACE) Score Index at Weeks 24 and 52
Description: GRACE index is a composite PsA disease activity score converted from AMDF, which was derived from TJC (0-68) and SJC (0-66), HAQ-DI (0-3), patient's global assessment of disease activity on arthritis and psoriasis (0-100 mm, 0=excellent and 100= poor), patient's assessment of skin disease activity (0-100 mm, 0=excellent and 100=poor), patient's global assessment of disease activity on arthritis (0-100 mm, 0=excellent and 100=poor), PASI (0-72), and PsA Quality of Life Index (derived as PsAQOL =25.355 + [2.367*HAQ-DI] - [0.234*SF-PCS] - [0.244*SF-MCS]), where HAQ-DI: HAQ-DI score (0-3, 0=least difficulty and 3=extreme difficulty), SF-PCS (Score ranges from 0 to 100, higher scores= better quality of life) and SF-MCS (score ranges from 0 to 100, higher scores= better quality of life). The total score is from 0-10, where lower score indicates better response. Higher score indicates more active disease activity. Negative change from baseline indicates improvement of PsA disease activity.
Time Frame: Baseline, Weeks 24 and 52
Population: as for outcome 63
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 114 | 123 | 125
units on a scale
  Week 24: number analyzed (Participants) | 113 | 121 | 124
  Week 24 | -0.998 (1.4808) | -2.493 (1.5195) | -2.751 (1.5060)
  Week 52: number analyzed (Participants) | 103 | 110 | 123
  Week 52 | -2.829 (1.5773) | -3.112 (1.7479) | -3.364 (1.4638)

84. Secondary Outcome: Change From Baseline in Psoriatic Arthritis Disease Activity (PASDAS) Score at Weeks 24 and 52
Description: as for outcome 33
Time Frame: Baseline, Weeks 24 and 52
Population: as for outcome 63
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 114 | 123 | 125
units on a scale
  Week 24: number analyzed (Participants) | 113 | 121 | 124
  Week 24 | -1.140 (1.4036) | -2.246 (1.4978) | -2.413 (1.3906)
  Week 52: number analyzed (Participants) | 103 | 110 | 123
  Week 52 | -2.748 (1.4706) | -2.897 (1.6788) | -3.026 (1.4446)

85. Secondary Outcome: Percentage of Participants Who Maintained an ACR 20 Response at Week 52 Among Participants Who Achieved an ACR 20 Response at Week 24
Description: as for outcome 15
Time Frame: Week 52
Population: FAS2 among participants achieved ACR20 response at Week 24. Here, N (number of participants analyzed) signifies number of participants analyzed for this OM. OM was planned to assess maintenance of guselkumab effect only through Week 52, hence data is reported for guselkumab 100mg q8w and guselkumab 100mg q4w arms only and not for placebo arm.
Measure: Number; unit: percentage of participants
Arm/Group | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 61 | 76
percentage of participants | 88.5 | 90.8

86. Secondary Outcome: Percentage of Participants Who Maintained an ACR 50 Response at Week 52 Among Participants Who Achieved an ACR 50 Response at Week 24
Description: as for outcome 16
Time Frame: Week 52
Population: FAS2 among participants achieved ACR50 response at Week 24. Here, N (number of participants analyzed) signifies number of participants analyzed for this OM. The OM was planned to assess maintenance of guselkumab effect only through Week 52, hence data is reported for guselkumab 100 mg q8w and guselkumab 100 mg q4w arms only and not for placebo arm.
Measure: Number; unit: percentage of participants
Arm/Group | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 37 | 46
percentage of participants | 83.8 | 91.3

87. Secondary Outcome: Percentage of Participants Who Maintained an ACR 70 Response at Week 52 Among Participants Who Achieved an ACR 70 Response at Week 24
Description: as for outcome 17
Time Frame: Week 52
Population: Analysis population is FAS2 among participants who achieved ACR 70 response at Week 24. The outcome measure was planned to assess the maintenance of guselkumab effect only through Week 52, hence the data in this outcome measure is reported for guselkumab 100 mg q8w and guselkumab 100 mg q4w arms only and not for placebo arm.
Measure: Number; unit: percentage of participants
Arm/Group | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 15 | 26
percentage of participants | 80.0 | 84.6

88. Secondary Outcome: Percentage of Participants Who Achieved >= 20%, >=50%, >=70%, and >=90% Improvement From Baseline in BASDAI Score at Weeks 24 and 52 Among Participants With Spondylitis and Peripheral Arthritis as Their Primary Arthritic Presentation of PsA
Description: as for outcome 37
Time Frame: Weeks 24 and 52
Population: Analysis population is FAS2 among the participants with spondylitis and peripheral arthritis and BASDAI score >0 at baseline. Here, n (number analyzed) signifies the number of participants analyzed at specified timepoints.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 21 | 24 | 20
percentage of participants
  Week 24: Participants with >=20% Improvement | 38.1 | 70.8 | 65.0
  Week 52: Participants with >=20% Improvement: number analyzed (Participants) | 21 | 22 | 20
  Week 52: Participants with >=20% Improvement | 66.7 | 72.7 | 85.0
  Week 24: Participants with >=50% Improvement | 19.0 | 41.7 | 35.0
  Week 52: Participants with >=50% Improvement | 52.4 | 59.1 | 50.0
  Week 24: Participants with >=70% Improvement | 14.3 | 29.2 | 5.0
  Week 52: Participants with >=70% Improvement | 28.6 | 40.9 | 20.0
  Week 24: Participants with >=90% Improvement | 0 | 16.7 | 0
  Week 52: Participants with >=90% Improvement | 9.5 | 13.6 | 15.0

89. Secondary Outcome: Percentage of Participants With Resolution of Enthesitis at Weeks 24, 36, 44 and 52 Among the Participants With Enthesitis at Baseline
Description: as for outcome 29
Time Frame: Weeks 24, 36, 44 and 52
Population: Analysis population is FAS2 among the participants with enthesitis (LEI) at baseline who achieved resolution of enthesitis at Week 24. Here, N (number of participants analyzed) signifies the number of participants analyzed for this outcome measure and n (number analyzed) signifies the number of participants analyzed at specified timepoints.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 71 | 71 | 71
percentage of participants
  Week 24 | 31.0 | 40.8 | 49.3
  Week 36: number analyzed (Participants) | 69 | 70 | 69
  Week 36 | 49.3 | 52.9 | 58.0
  Week 44: number analyzed (Participants) | 67 | 69 | 71
  Week 44 | 58.2 | 46.4 | 71.8
  Week 52: number analyzed (Participants) | 63 | 64 | 70
  Week 52 | 69.8 | 56.3 | 62.9

90. Secondary Outcome: Percentage of Participants With Resolution of Dactylitis at Weeks 24, 36, 44 and 52 Among Participants With Dactylitis at Baseline
Description: as for outcome 13
Time Frame: Weeks 24, 36, 44 and 52
Population: Analysis population is FAS2 among the participants with dactylitis at baseline. Here, n (number analyzed) signifies the number of participants analyzed at specified timepoints.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 47 | 49 | 37
percentage of participants
  Week 24 | 61.7 | 67.3 | 64.9
  Week 36: number analyzed (Participants) | 44 | 46 | 35
  Week 36 | 79.5 | 67.4 | 82.9
  Week 44: number analyzed (Participants) | 46 | 46 | 37
  Week 44 | 84.8 | 76.1 | 83.8
  Week 52: number analyzed (Participants) | 43 | 44 | 37
  Week 52 | 81.4 | 79.5 | 78.4

91. Secondary Outcome: Change From Baseline in Enthesitis Score (Based on SPARCC) at Weeks 24, 36, 44 and 52 Among the Participants With Enthesitis at Baseline
Description: Enthesitis was assessed using the Spondyloarthritis Research Consortium of Canada (SPARCC). The SPARCC developed a measure for enthesitis in general spondyloarthritis which evaluates the presence or absence of pain by applying local pressure to the following entheses: supraspinatus insertion (left and right), medial epicondyle humerus (left and right), lateral epicondyle humerus (left and right), greater trochanter (left and right), quadriceps-to-patella (left and right), patellar-tibia (left and right), achilles tendon insertion (left and right), plantar fascia (left and right). Tenderness on examination was recorded as either present (1) or absent (0) for each of the 16 sites for an overall score range of 0-16. Higher scores indicate more severe enthesitis. Negative changes from baseline indicate improvement of enthesitis.
Time Frame: Baseline, Weeks 24, 36, 44 and 52
Population: Analysis population is FAS2 among the participants with enthesitis (SPARCC) at baseline. Here, n (number analyzed) signifies the number of participants analyzed at specified timepoints.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 77 | 85 | 82
units on a scale
  Week 24 | -1.9 (3.55) | -2.7 (3.68) | -3.0 (3.60)
  Week 36: number analyzed (Participants) | 73 | 83 | 80
  Week 36 | -3.1 (3.61) | -3.4 (3.90) | -3.6 (3.52)
  Week 44: number analyzed (Participants) | 71 | 82 | 82
  Week 44 | -3.6 (3.67) | -3.6 (3.82) | -4.1 (3.55)
  Week 52: number analyzed (Participants) | 69 | 76 | 81
  Week 52 | -3.9 (3.57) | -4.1 (4.04) | -4.0 (3.51)

92. Secondary Outcome: Change From Baseline in Enthesitis Score (Based on LEI) at Weeks 24, 36, 44 and 52 Among the Participants With Enthesitis at Baseline
Description: as for outcome 30
Time Frame: Baseline, Weeks 24, 36, 44 and 52
Population: Analysis population is FAS2 among the participants with enthesitis (LEI) at baseline. Here, N (number of participants analyzed) signifies the number of participants analyzed for this outcome measure and n (number analyzed) signifies the number of participants analyzed at specified timepoints.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 71 | 71 | 71
units on a scale
  Week 24 | -1.0 (1.68) | -1.2 (1.95) | -1.8 (1.93)
  Week 36: number analyzed (Participants) | 69 | 70 | 69
  Week 36 | -1.4 (1.73) | -1.3 (2.04) | -2.0 (1.68)
  Week 44: number analyzed (Participants) | 67 | 69 | 71
  Week 44 | -1.6 (1.90) | -1.6 (1.70) | -2.4 (1.68)
  Week 52: number analyzed (Participants) | 63 | 64 | 70
  Week 52 | -1.9 (1.65) | -1.8 (1.66) | -2.0 (1.87)

93. Secondary Outcome: Change From Baseline in Dactylitis Score at Weeks 24, 36, 44 and 52 Among the Participants With Dactylitis at Baseline
Description: as for outcome 32
Time Frame: Baseline, Weeks 24, 36, 44 and 52
Population: as for outcome 90
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 47 | 49 | 37
units on a scale
  Week 24 | -4.0 (6.08) | -6.2 (10.31) | -6.6 (11.08)
  Week 36: number analyzed (Participants) | 44 | 46 | 35
  Week 36 | -6.0 (7.17) | -6.4 (10.91) | -7.7 (11.58)
  Week 44: number analyzed (Participants) | 46 | 46 | 37
  Week 44 | -5.3 (5.61) | -7.2 (10.57) | -7.5 (11.41)
  Week 52: number analyzed (Participants) | 43 | 44 | 37
  Week 52 | -5.7 (5.86) | -7.8 (10.55) | -7.6 (10.91)

94. Secondary Outcome: Percentage of Participants With an IGA Score of 0 (Cleared) or 1 (Cleared) at Weeks 24 and 52 Among Participants With >=3% BSA Psoriatic Involvement and an IGA Score of >=2 at Baseline
Description: A psoriasis IGA response was defined as an IGA score of 0 (cleared) or 1 (minimal) and >= 2 grade reduction from baseline in the IGA psoriasis score. The IGA documents the investigator's assessment of the patient's psoriasis and lesions are graded for induration, erythema and scaling, each using a 5 point scale: 0 (no evidence), 1 (minimal), 2 (mild), 3 (moderate), and 4 (severe). The IGA score of psoriasis was based upon the average of induration, erythema and scaling scores. The participant's psoriasis was assessed as cleared (0), minimal (1), mild (2), moderate (3), or severe (4).
Time Frame: Weeks 24 and 52
Population: as for outcome 74
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 68 | 82 | 88
percentage of participants
  Week 24: number analyzed (Participants) | 68 | 81 | 88
  Week 24 | 8.8 | 38.3 | 54.5
  Week 52: number analyzed (Participants) | 65 | 75 | 88
  Week 52 | 66.2 | 53.3 | 67.0

95. Secondary Outcome: Change From Baseline in SF-36 Physical Component Summary (PCS) Score at Weeks 24, 36 and 52
Description: as for outcome 9
Time Frame: Baseline, Weeks 24, 36 and 52
Population: as for outcome 63
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 114 | 123 | 125
units on a scale
  Week 24: number analyzed (Participants) | 114 | 123 | 124
  Week 24 | 2.700 (7.1649) | 6.505 (7.7137) | 6.560 (7.7566)
  Week 36: number analyzed (Participants) | 107 | 119 | 120
  Week 36 | 5.456 (8.0353) | 7.439 (8.5626) | 7.162 (7.9890)
  Week 52: number analyzed (Participants) | 104 | 114 | 124
  Week 52 | 6.905 (7.9376) | 7.278 (8.0648) | 8.517 (8.2717)

96. Secondary Outcome: Change From Baseline in SF-36 Mental Component Summary (MCS) Score at Weeks 24, 36 and 52
Description: as for outcome 12
Time Frame: Baseline, Weeks 24, 36 and 52
Population: as for outcome 63
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 114 | 123 | 125
units on a scale
  Week 24: number analyzed (Participants) | 114 | 123 | 124
  Week 24 | 1.827 (8.1508) | 3.027 (10.6157) | 3.796 (8.7396)
  Week 36: number analyzed (Participants) | 107 | 119 | 120
  Week 36 | 3.612 (7.2322) | 4.300 (10.2373) | 4.326 (9.2709)
  Week 52: number analyzed (Participants) | 104 | 114 | 124
  Week 52 | 4.240 (8.1200) | 5.139 (9.1719) | 4.931 (8.9482)

97. Secondary Outcome: Change From Baseline in Norm Based Scores of SF-36 Scales at Week 24, 36 and 52
Description: as for outcome 52
Time Frame: Baseline, Weeks 24, 36 and 52
Population: Analysis population is FAS2. Here, n (number analyzed) signifies the number of participants analyzed at specified timepoints for specific categories.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 114 | 123 | 125
units on a scale
  Week 24: Physical Functioning: number analyzed (Participants) | 114 | 123 | 124
  Week 24: Physical Functioning | 1.914 (8.8644) | 6.006 (7.9608) | 6.652 (8.4730)
  Week 36: Physical Functioning: number analyzed (Participants) | 107 | 119 | 120
  Week 36: Physical Functioning | 5.008 (8.6461) | 6.900 (8.5458) | 7.114 (8.8941)
  Week 52: Physical Functioning: number analyzed (Participants) | 104 | 114 | 124
  Week 52: Physical Functioning | 6.257 (8.3753) | 7.000 (8.0953) | 8.720 (8.9738)
  Week 24: Role-physical: number analyzed (Participants) | 114 | 123 | 124
  Week 24: Role-physical | 3.053 (7.6460) | 5.239 (8.2864) | 5.215 (7.5241)
  Week 36: Role-physical: number analyzed (Participants) | 107 | 119 | 120
  Week 36: Role-physical | 4.701 (8.1572) | 6.245 (7.8346) | 6.250 (7.9040)
  Week 52: Role-physical: number analyzed (Participants) | 104 | 114 | 124
  Week 52: Role-physical | 5.873 (8.8847) | 6.126 (8.1008) | 7.063 (8.2579)
  Week 24: Bodily Pain: number analyzed (Participants) | 114 | 123 | 124
  Week 24: Bodily Pain | 3.388 (7.2056) | 7.058 (8.8315) | 7.215 (9.1129)
  Week 36: Bodily Pain: number analyzed (Participants) | 107 | 119 | 120
  Week 36: Bodily Pain | 6.477 (8.6363) | 8.487 (8.8135) | 7.348 (9.0965)
  Week 52: Bodily Pain: number analyzed (Participants) | 104 | 114 | 124
  Week 52: Bodily Pain | 8.331 (8.1585) | 8.781 (8.5691) | 8.958 (9.1783)
  Week 24: General Health: number analyzed (Participants) | 114 | 123 | 124
  Week 24: General Health | 1.819 (6.9497) | 4.361 (7.5573) | 5.066 (7.1334)
  Week 36: General Health: number analyzed (Participants) | 107 | 119 | 120
  Week 36: General Health | 3.742 (8.2079) | 5.638 (8.4919) | 5.540 (7.4840)
  Week 52: General Health: number analyzed (Participants) | 104 | 123 | 125
  Week 52: General Health | 4.677 (7.8944) | 5.547 (7.8712) | 6.442 (7.9374)
  Week 24: Vitality: number analyzed (Participants) | 114 | 123 | 124
  Week 24: Vitality | 2.684 (9.0049) | 5.652 (9.6943) | 6.158 (7.8842)
  Week 36: Vitality: number analyzed (Participants) | 107 | 119 | 120
  Week 36: Vitality | 6.303 (9.0307) | 7.065 (8.6659) | 7.353 (8.7656)
  Week 52: Vitality: number analyzed (Participants) | 104 | 114 | 124
  Week 52: Vitality | 7.742 (8.7476) | 7.558 (9.1600) | 8.218 (8.5308)
  Week 24: Social Function | 2.419 (8.8289) | 5.666 (9.3449) | 4.932 (9.5887)
  Week 36: Social Function: number analyzed (Participants) | 107 | 119 | 120
  Week 36: Social Function | 4.873 (9.1477) | 5.899 (9.9762) | 5.598 (10.5240)
  Week 52: Social Function: number analyzed (Participants) | 104 | 114 | 124
  Week 52: Social Function | 5.351 (8.9264) | 6.729 (8.4844) | 6.428 (10.1397)
  Week 24: Role-emotional: number analyzed (Participants) | 114 | 123 | 124
  Week 24: Role-emotional | 1.833 (9.0800) | 2.265 (10.6155) | 3.706 (9.3529)
  Week 36: Role-emotional: number analyzed (Participants) | 107 | 119 | 120
  Week 36: Role-emotional | 3.580 (8.5353) | 4.301 (10.1127) | 3.685 (10.5307)
  Week 52: Role-emotional: number analyzed (Participants) | 104 | 114 | 124
  Week 52: Role-emotional | 4.520 (8.8658) | 4.979 (10.2956) | 4.830 (9.9053)
  Week 24: Mental Health: number analyzed (Participants) | 114 | 123 | 124
  Week 24: Mental Health | 1.905 (8.1196) | 4.062 (10.0610) | 4.873 (8.6431)
  Week 36: Mental Health: number analyzed (Participants) | 107 | 119 | 120
  Week 36: Mental Health | 3.472 (7.0761) | 5.056 (9.7930) | 5.559 (8.9957)
  Week 52: Mental Health: number analyzed (Participants) | 104 | 114 | 124
  Week 52: Mental Health | 4.251 (8.3059) | 5.553 (8.4255) | 6.223 (8.8360)

98. Secondary Outcome: Change From Baseline in Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue Score at Weeks 24, 36 and 52
Description: as for outcome 55
Time Frame: Baseline, Weeks 24, 36 and 52
Population: as for outcome 63
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 114 | 123 | 125
units on a scale
  Week 24 | 2.605 (8.3142) | 5.862 (10.3941) | 5.576 (7.7670)
  Week 36: number analyzed (Participants) | 107 | 119 | 121
  Week 36 | 5.981 (8.3846) | 7.252 (9.7182) | 5.917 (8.5123)
  Week 52: number analyzed (Participants) | 104 | 114 | 124
  Week 52 | 6.577 (9.4105) | 7.482 (9.6342) | 6.911 (8.3986)

99. Secondary Outcome: Percentage of Participants Who Achieved >=4-point Improvement From Baseline in FACIT-Fatigue Score at Weeks 24, 36 and 52
Description: as for outcome 55
Time Frame: Weeks 24, 36 and 52
Population: as for outcome 63
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 114 | 123 | 125
percentage of participants
  Week 24 | 41.2 | 55.3 | 64.8
  Week 36: number analyzed (Participants) | 107 | 119 | 121
  Week 36 | 60.7 | 58.0 | 66.1
  Week 52: number analyzed (Participants) | 104 | 114 | 124
  Week 52 | 63.5 | 61.4 | 63.7

100. Secondary Outcome: Change From Baseline in Patient-Reported Outcomes Measurement Information System (PROMIS)-29 Scores at Weeks 24, 36 and 52
Description: as for outcome 60
Time Frame: Baseline, Weeks 24, 36 and 52
Population: as for outcome 63
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Placebo | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 114 | 123 | 125
T-score
  Week 24: Anxiety Score | -1.482 (8.3526) | -3.680 (9.8122) | -3.115 (7.9491)
  Week 36: Anxiety Score: number analyzed (Participants) | 107 | 119 | 121
  Week 36: Anxiety Score | -2.410 (7.6503) | -3.929 (8.9614) | -2.961 (8.4679)
  Week 52: Anxiety Score: number analyzed (Participants) | 104 | 114 | 124
  Week 52: Anxiety Score | -3.640 (8.3601) | -4.279 (9.6488) | -3.075 (8.5784)
  Week 24: Depression Score | -0.601 (8.3133) | -3.963 (8.5473) | -2.706 (8.1872)
  Week 36: Depression Score: number analyzed (Participants) | 107 | 119 | 121
  Week 36: Depression Score | -0.933 (7.1629) | -3.916 (8.6211) | -2.987 (7.8786)
  Week 52: Depression Score: number analyzed (Participants) | 104 | 114 | 124
  Week 52: Depression Score | -2.488 (7.8259) | -4.004 (7.5271) | -2.985 (8.0519)
  Week 24: Fatigue Score | -2.104 (7.5625) | -4.780 (9.7044) | -4.757 (7.7779)
  Week 36: Fatigue Score: number analyzed (Participants) | 107 | 119 | 121
  Week 36: Fatigue Score | -5.533 (8.3256) | -5.857 (8.8525) | -5.693 (9.3854)
  Week 52: Fatigue Score: number analyzed (Participants) | 104 | 114 | 124
  Week 52: Fatigue Score | -5.720 (9.0165) | -6.773 (8.5608) | -5.583 (8.1099)
  Week 24: Pain Interference Score | -2.811 (5.9890) | -5.810 (7.5201) | -5.423 (7.1593)
  Week 36: Pain Interference Score: number analyzed (Participants) | 107 | 119 | 121
  Week 36: Pain Interference Score | -5.344 (7.2500) | -6.754 (8.0520) | -5.882 (7.5121)
  Week 52: Pain Interference Score: number analyzed (Participants) | 104 | 114 | 124
  Week 52: Pain Interference Score | -6.334 (6.9940) | -6.972 (8.2440) | -6.242 (7.4767)
  Week 24: Physical Function Score | 1.682 (5.9909) | 4.101 (7.1353) | 5.030 (6.5259)
  Week 36: Physical Function Score: number analyzed (Participants) | 107 | 119 | 121
  Week 36: Physical Function Score | 3.093 (6.5712) | 4.970 (7.0012) | 5.264 (7.0643)
  Week 52: Physical Function Score: number analyzed (Participants) | 104 | 114 | 124
  Week 52: Physical Function Score | 4.245 (6.1363) | 5.033 (7.0184) | 5.920 (6.9852)
  Week 24: Sleep Disturbance Score | -1.497 (5.7591) | -3.750 (6.8758) | -2.549 (6.7263)
  Week 36: Sleep Disturbance Score: number analyzed (Participants) | 107 | 119 | 121
  Week 36: Sleep Disturbance Score | -2.767 (5.7630) | -3.853 (6.5505) | -4.096 (6.8724)
  Week 52: Sleep Disturbance Score: number analyzed (Participants) | 104 | 114 | 124
  Week 52: Sleep Disturbance Score | -3.290 (5.8368) | -4.375 (6.5738) | -3.856 (6.1181)
  Week24:Satisfaction-Social Role and Activity Score | 1.666 (7.2572) | 5.308 (8.5808) | 4.235 (7.4745)
  Week36:Satisfaction-Social Role and Activity Score: number analyzed (Participants) | 107 | 119 | 121
  Week36:Satisfaction-Social Role and Activity Score | 4.120 (8.1899) | 6.270 (8.8798) | 4.517 (7.9605)
  Week52:Satisfaction-Social Role and Activity Score: number analyzed (Participants) | 104 | 114 | 124
  Week52:Satisfaction-Social Role and Activity Score | 4.885 (8.7421) | 6.607 (7.8438) | 5.347 (8.1806)
  Week 24: Pain Intensity Score | -0.737 (2.0911) | -2.098 (2.4104) | -2.320 (2.4449)
  Week 36: Pain Intensity Score: number analyzed (Participants) | 107 | 119 | 121
  Week 36: Pain Intensity Score | -1.720 (2.3424) | -2.496 (2.4212) | -2.488 (2.4018)
  Week 52: Pain Intensity Score: number analyzed (Participants) | 104 | 114 | 124
  Week 52: Pain Intensity Score | -2.462 (2.3480) | -2.711 (2.4844) | -2.847 (2.5377)

ADVERSE EVENTS:
Time Frame: Up to Week 60
Description: Safety analysis set included participants who were randomized at Week 0 and received at least 1 (partial or complete) administration of study agent and were analyzed according to the actual treatment received after randomization. Data for Guselkumab 100 mg q8w and q4w arms was planned to be reported separately for Week 0 to 24 and Week 0 to 60.
Groups:
- Placebo (CP): Participants received placebo matched to guselkumab subcutaneous injections every 4 weeks through Week 20 in the placebo controlled period (CP). Data prior to the first administration of guselkumab, or through the last follow-up visit if the participant did not receive any guselkumab, were included.
- Guselkumab 100 mg q8w (CP): Participants received guselkumab 100 mg subcutaneous injections at Weeks 0 and 4, then every 8 weeks and placebo matched to guselkumab injections at other visits through Week 20 in the placebo controlled period (CP). Data through Week 24, or through the last follow-up visit if the participant did not receive any study drug at or after Week 24, were included.
- Guselkumab 100 mg q4w (CP): Participants received guselkumab 100 mg subcutaneous injections every 4 weeks from Week 0 through Week 20 in the placebo controlled period (CP). Data through Week 24, or through the last follow-up visit if the participant did not receive any study drug at or after Week 24, were included.
- Placebo to Guselkumab 100 mg q4w (ACP Through Week 60): Participants who received placebo matched to guselkumab subcutaneous injections every 4 weeks through Week 20 in the placebo controlled period (CP) received guselkumab 100 mg subcutaneous injections every 4 weeks from Week 24 through Week 48. Data from the first administration of guselkumab through Week 60 were included.
- Guselkumab 100 mg q8w (Through Week 60): Participants received guselkumab 100 mg subcutaneous injections at Weeks 0 and 4, then every 8 weeks and placebo matched to guselkumab injections at other visits through Week 48. Data from Week 0 through Week 60 were included.
- Guselkumab 100 mg q4w (Through Week 60): Participants received guselkumab 100 mg subcutaneous injections every 4 weeks from Week 0 through Week 48. Data from Week 0 through Week 60 were included.
Arm/Group | Placebo (CP) | Guselkumab 100 mg q8w (CP) | Guselkumab 100 mg q4w (CP) | Placebo to Guselkumab 100 mg q4w (ACP Through Week 60) | Guselkumab 100 mg q8w (Through Week 60) | Guselkumab 100 mg q4w (Through Week 60)
All-Cause Mortality (participants affected / at risk) | 2/126 | 0/127 | 0/128 | 0/114 | 0/127 | 0/128
Serious Adverse Events (participants affected / at risk) | 5/126 | 4/127 | 0/128 | 4/114 | 8/127 | 4/128
Other Adverse Events (participants affected / at risk) | 25/126 | 38/127 | 28/128 | 25/114 | 48/127 | 41/128
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (CP) (N=126) | Guselkumab 100 mg q8w (CP) (N=127) | Guselkumab 100 mg q4w (CP) (N=128) | Placebo to Guselkumab 100 mg q4w (ACP Through Week 60) (N=114) | Guselkumab 100 mg q8w (Through Week 60) (N=127) | Guselkumab 100 mg q4w (Through Week 60) (N=128)
Arrhythmia Supraventricular (Cardiac disorders) | 0 | 1 | 0 | 0 | 1 | 0
Atrial Fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Cardiac Failure (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Mechanical Ileus (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0
Pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Abscess Limb (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Urosepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Hand Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Head Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Meniscus Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Foot Deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Lumbar Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Plasma Cell Myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 1 | 0
Renal Colic (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Breast Enlargement (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cervical Dysplasia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 1 | 0
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pustular Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Venous Thrombosis Limb (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (CP) (N=126) | Guselkumab 100 mg q8w (CP) (N=127) | Guselkumab 100 mg q4w (CP) (N=128) | Placebo to Guselkumab 100 mg q4w (ACP Through Week 60) (N=114) | Guselkumab 100 mg q8w (Through Week 60) (N=127) | Guselkumab 100 mg q4w (Through Week 60) (N=128)
Bronchitis (Infections and infestations) | 1 | 5 | 1 | 3 | 9 | 2
Nasopharyngitis (Infections and infestations) | 8 | 16 | 7 | 13 | 21 | 14
Upper Respiratory Tract Infection (Infections and infestations) | 8 | 7 | 11 | 8 | 10 | 16
Alanine Aminotransferase Increased (Investigations) | 3 | 8 | 5 | 4 | 9 | 9
Aspartate Aminotransferase Increased (Investigations) | 3 | 9 | 3 | 4 | 11 | 6
Enthesopathy (Musculoskeletal and connective tissue disorders) | 6 | 6 | 6 | 0 | 7 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2018-01-25): https://cdn.clinicaltrials.gov/large-docs/96/NCT03162796/Prot_000.pdf
  • Statistical Analysis Plan (2019-03-21): https://cdn.clinicaltrials.gov/large-docs/96/NCT03162796/SAP_001.pdf